CLINICAL TRIAL: NCT04047862
Title: Phase 1/1b Study Investigating Safety, Tolerability, PK and Antitumor Activity of Anti-TIGIT Monoclonal Antibody BGB-A1217 in Combination With Anti-PD-1 Monoclonal Antibody Tislelizumab in Patients With Advanced Solid Tumors
Brief Title: Study of Ociperlimab (BGB-A1217) in Combination With Tislelizumab in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-900-105; AdvanTIG-105 (Other: BeiGene); CTR20202608 (Other: ChinaDrugTrials)
Record Dates: First submitted 2019-08-01; First posted 2019-08-07 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Locally Advanced and Metastatic Solid Tumors
Keywords: BGB-A1217; Anti-TIGIT antibody; Tislelizumab; anti-PD-1 antibody; Ociperlimab
MeSH Terms: interventions — tislelizumab; Pemetrexed; Paclitaxel; Taxes; Carboplatin; Cisplatin; Etoposide; Fluorouracil; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (19):
- Phase 1: Dose Escalation: Ociperlimab 50 mg + Tislelizumab 200 mg (Experimental): Participants received ociperlimab 50 milligrams (mg) intravenous (IV) infusion on Day 1 of each cycle (cycle 1= 28 days) and tislelizumab 200 mg IV infusion on Day 8 of Cycle 1. If tolerated, participants received ociperlimab and tislelizumab doses IV on Cycle 2 Day 1 (cycle 2 onwards = 21 days) and thereafter every 21 days (that is, [i.e.], every 3 weeks [Q3W]) until disease progression, adverse events (AEs), participant withdrew consent, lost to follow-up or death, whichever came first.
  Interventions: Drug: Ociperlimab; Drug: Tislelizumab
- Phase 1: Dose Escalation: Ociperlimab 150 mg + Tislelizumab 200 mg (Experimental): Participants received ociperlimab 150 mg IV infusion on Day 1 of each cycle (cycle 1= 28 days) and tislelizumab 200 mg IV infusion on Day 8 of Cycle 1. If tolerated, participants received ociperlimab and tislelizumab doses IV on Cycle 2 Day 1 (cycle 2 onwards = 21 days) and thereafter every 21 days (i.e. Q3W) until disease progression, intolerable toxicity, or withdrawal of consent.
  Interventions: Drug: Ociperlimab; Drug: Tislelizumab
- Phase 1: Dose Escalation: Ociperlimab 450 mg + Tislelizumab 200 mg (Experimental): Participants received ociperlimab 450 mg IV infusion on Day 1 of each cycle (cycle 1= 28 days) and tislelizumab 200 mg IV infusion on Day 8 of Cycle 1. If tolerated, participants received ociperlimab and tislelizumab doses IV on Cycle 2 Day 1 (cycle 2 onwards = 21 days) and thereafter every 21 days (i.e. Q3W) until disease progression, intolerable toxicity, or withdrawal of consent.
  Interventions: Drug: Ociperlimab; Drug: Tislelizumab
- Phase 1: Dose Escalation: Ociperlimab 900 mg + Tislelizumab 200 mg (Experimental): Participants received ociperlimab 900 mg IV infusion on Day 1 of each cycle (cycle 1= 28 days) and tislelizumab 200 mg IV infusion on Day 8 of Cycle 1. If tolerated, participants received ociperlimab and tislelizumab doses IV on Cycle 2 Day 1 (cycle 2 onwards = 21 days) and thereafter every 21 days (i.e. Q3W) until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
  Interventions: Drug: Ociperlimab; Drug: Tislelizumab
- Phase 1: Dose Escalation: Ociperlimab 1800 mg + Tislelizumab 200 mg (Experimental): Participants received ociperlimab 1800 mg IV infusion on Day 1 of each cycle (cycle 1= 28 days) and tislelizumab 200 mg IV infusion on Day 8 of Cycle 1. If tolerated, participants received ociperlimab and tislelizumab doses IV on Cycle 2 Day 1 (cycle 2 onwards = 21 days) and thereafter every 21 days (i.e. Q3W) until disease progression, intolerable toxicity, or withdrawal of consent.
  Interventions: Drug: Ociperlimab; Drug: Tislelizumab
- Phase 1: Dose Verification: Cohort 1A (Ociperlimab 900 mg) (Experimental): Participants received ociperlimab 900 mg as monotherapy IV infusion on Day 1 of each 21-day treatment cycle until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
  Interventions: Drug: Ociperlimab
- Phase 1: Dose Verification: Cohort 1B (Ociperlimab 900 mg + Tislelizumab 200 mg) (Experimental): Participants received ociperlimab 900 mg as IV infusion on Day 1 of each 21-day treatment cycle and tislelizumab 200 mg IV infusion once every 21 days (i.e. Q3W) until disease progression, intolerable toxicity, or withdrawal of consent.
  Interventions: Drug: Ociperlimab; Drug: Tislelizumab
- Phase 1b: Dose Expansion: Cohort 1 (Experimental): Participants with metastatic squamous non-small cell lung cancer (NSCLC) received treatment with ociperlimab 900 mg IV infusion along with tislelizumab 200 mg IV infusion on Day 1 of each 21-day cycle. Participants also received 4 to 6 cycles of chemotherapy with carboplatin at an area under the curve (AUC) 5 or 6 (Day 1) + paclitaxel 200 or 175 mg/m^2 (Day 1) or nab paclitaxel 100 mg/m^2 (Days 1, 8 and 15) Q3W p until disease progression, intolerable toxicity, or withdrawal of consent.
  Interventions: Drug: Ociperlimab; Drug: Tislelizumab; Drug: Paclitaxel; Drug: Nab paclitaxel; Drug: Carboplatin
- Phase 1b: Dose Expansion: Cohort 2 (Experimental): Participants with metastatic non-squamous NSCLC received treatment with ociperlimab 900 mg IV infusion and tislelizumab 200 mg IV infusion on Day 1 of each 21-day cycle. Participants also received cisplatin 75 mg/m^2 or carboplatin (AUC 5) and pemetrexed 500 mg/m^2 (on Day 1) Q3W for 4-6 cycles followed by ociperlimab 900 mg + tislelizumab 200 mg + pemetrexed 500 mg/m^2 on Day 1 Q3W until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
  Interventions: Drug: Ociperlimab; Drug: Tislelizumab; Drug: Pemetrexed; Drug: Carboplatin; Drug: Cisplatin
- Phase 1b: Dose Expansion: Cohort 3 (Experimental): Participants with metastatic NSCLC (programmed cell death protein-ligand 1 [PD-L1] positive, tumor cell [TC] >=1%) were treated with ociperlimab 900 mg IV infusion and tislelizumab 200 mg IV infusion on Day 1 of each 21-day cycle until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
  Interventions: Drug: Ociperlimab; Drug: Tislelizumab
- Phase 1b: Dose Expansion: Cohort 4 (Experimental): Participants with extensive-stage small-cell lung cancer (SCLC) received treatment with ociperlimab 900 mg IV infusion, tislelizumab 200 mg IV infusion. Participants also received 4 cycles of etoposide 100 mg/m^2 (on Days 1, 2, 3), and cisplatin 75 mg/m^2 or carboplatin AUC 5 (Day 1) Q3W, followed by ociperlimab 900 mg (Day 1) + tislelizumab 200 mg (Day 1) Q3W until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
  Interventions: Drug: Ociperlimab; Drug: Tislelizumab; Drug: Carboplatin; Drug: Cisplatin; Drug: Etoposide
- Phase 1b: Dose Expansion: Cohort 5 (Experimental): Checkpoint inhibitor (CPI)-experienced NSCLC participants received treatment with ociperlimab 900 mg IV infusion and tislelizumab 200 mg IV infusions on Day 1 of each 21-day cycle until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
  Interventions: Drug: Ociperlimab; Drug: Tislelizumab
- Phase 1b: Dose Expansion: Cohort 6 (Experimental): Participants with metastatic esophageal squamous cell carcinoma (ESCC) received treatment with 6 cycles of ociperlimab 900 mg (Day 1) IV infusion, tislelizumab 200 mg (Day 1) IV infusion, cisplatin 75 mg/m^2 (Day 1), and 5-fluorouracil 750-800 mg/m^2 (5-FU; Day 1 to Day 5) or paclitaxel 200 or 175 mg/m^2 (Day 1) Q3W followed by ociperlimab 900 mg and tislelizumab 200 mg on Day 1 of every 21-day cycle until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
  Interventions: Drug: Ociperlimab; Drug: Tislelizumab; Drug: Paclitaxel; Drug: Cisplatin; Drug: 5fluorouracil
- Phase 1b: Dose Expansion: Cohort 7 (Experimental): Participants with metastatic esophageal adenocarcinoma (EAC) received treatment with 6 cycles of ociperlimab 900 mg (Day 1) IV infusion, tislelizumab 200 mg (Day 1) IV infusion, cisplatin 75 mg/m^2 (Day 1), and 5-Fluorouracil 750-800 mg/m^2 (5-FU; Day 1 to Day 5) or paclitaxel 200 or 175 mg/m^2 (Day 1) Q3W followed by ociperlimab 900 mg and tislelizumab 200 mg on Day 1 of every 21-day cycle until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
  Interventions: Drug: Ociperlimab; Drug: Tislelizumab; Drug: Paclitaxel; Drug: Cisplatin; Drug: 5fluorouracil
- Phase 1b: Dose Expansion: Cohort 8 (Experimental): Participants with recurrent or metastatic head and neck squamous cell carcinoma (HNSCC; PD-L1 positive, visually estimated Combined Positive Score [vCPS] >= 1%) received treatment with ociperlimab 900 mg IV infusion and tislelizumab 200 mg IV infusions on Day 1 of every 21-day cycle until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
  Interventions: Drug: Ociperlimab; Drug: Tislelizumab
- Phase 1b: Dose Expansion: Cohort 9 (Experimental): Participants with unresectable, locally advanced, recurrent, or metastatic gastric or gastroesophageal junction (G/GEJ) adenocarcinoma received treatment with 6 cycles of ociperlimab 900 mg (Day 1) IV infusion, tislelizumab 200 mg (Day 1) IV infusion, (oxaliplatin 1300 mg/m^2 [Day 1] and capecitabine 1000 mg/m^2 [Day 1-14 twice daily]), or (cisplatin 75 mg/m^2 [Day], and 5-FU 750-800 mg/m^2 [Day 1-5]) Q3W followed by ociperlimab 900 mg (Day 1), tislelizumab 200 mg (Day 1) + capecitabine 1000 mg/m^2 twice daily (Day 1-14) Q3W until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
  Interventions: Drug: Ociperlimab; Drug: Tislelizumab; Drug: Cisplatin; Drug: 5fluorouracil; Drug: Oxaliplatin; Drug: Capecitabine
- Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 450 mg + Tislelizumab 200 mg) (Experimental): articipants with metastatic NSCLC (PD-L1 positive, TC >= 1%) received treatment with ociperlimab 450 mg IV infusion and tislelizumab 200 mg IV infusion on Day 1 of every 21-day cycle until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
  Interventions: Drug: Ociperlimab; Drug: Tislelizumab
- Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 900 mg + Tislelizumab 200 mg) (Experimental): Participants with metastatic NSCLC (PD-L1 positive, TC >= 1%) received treatment with ociperlimab 900 mg IV infusion and tislelizumab 200 mg IV infusion on Day 1 of every 21-day cycle until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
  Interventions: Drug: Ociperlimab; Drug: Tislelizumab
- Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 1800 mg + Tislelizumab 200 mg) (Experimental): Participants with metastatic NSCLC (PD-L1 positive, TC >= 1%) received treatment with ociperlimab 1800 mg IV infusion and tislelizumab 200 mg IV infusion on Day 1 of every 21-day cycle until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
  Interventions: Drug: Ociperlimab; Drug: Tislelizumab

INTERVENTIONS:
Drug: Ociperlimab — Administered as an intravenous (IV) injection
Drug: Tislelizumab — Administered as an IV injection
  Arms: Phase 1: Dose Escalation: Ociperlimab 150 mg + Tislelizumab 200 mg; Phase 1: Dose Escalation: Ociperlimab 1800 mg + Tislelizumab 200 mg; Phase 1: Dose Escalation: Ociperlimab 450 mg + Tislelizumab 200 mg; Phase 1: Dose Escalation: Ociperlimab 50 mg + Tislelizumab 200 mg; Phase 1: Dose Escalation: Ociperlimab 900 mg + Tislelizumab 200 mg; Phase 1: Dose Verification: Cohort 1B (Ociperlimab 900 mg + Tislelizumab 200 mg); Phase 1b: Dose Expansion: Cohort 1; Phase 1b: Dose Expansion: Cohort 2; Phase 1b: Dose Expansion: Cohort 3; Phase 1b: Dose Expansion: Cohort 4; Phase 1b: Dose Expansion: Cohort 5; Phase 1b: Dose Expansion: Cohort 6; Phase 1b: Dose Expansion: Cohort 7; Phase 1b: Dose Expansion: Cohort 8; Phase 1b: Dose Expansion: Cohort 9; Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 1800 mg + Tislelizumab 200 mg); Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 450 mg + Tislelizumab 200 mg); Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 900 mg + Tislelizumab 200 mg)
Drug: Pemetrexed — Administered in accordance with local guidelines, prescribing information/summary of product
  Arms: Phase 1b: Dose Expansion: Cohort 2
Drug: Paclitaxel — Administered in accordance with local guidelines , prescribing information/summary of product
  Arms: Phase 1b: Dose Expansion: Cohort 1; Phase 1b: Dose Expansion: Cohort 6; Phase 1b: Dose Expansion: Cohort 7
Drug: Nab paclitaxel — Administered in accordance with local guidelines , prescribing information/summary of product
  Arms: Phase 1b: Dose Expansion: Cohort 1
Drug: Carboplatin — Administered in accordance with local guidelines , prescribing information/summary of product
  Arms: Phase 1b: Dose Expansion: Cohort 1; Phase 1b: Dose Expansion: Cohort 2; Phase 1b: Dose Expansion: Cohort 4
Drug: Cisplatin — Administered in accordance with local guidelines , prescribing information/summary of product
  Arms: Phase 1b: Dose Expansion: Cohort 2; Phase 1b: Dose Expansion: Cohort 4; Phase 1b: Dose Expansion: Cohort 6; Phase 1b: Dose Expansion: Cohort 7; Phase 1b: Dose Expansion: Cohort 9
Drug: Etoposide — Administered in accordance with local guidelines , prescribing information/summary of product
  Arms: Phase 1b: Dose Expansion: Cohort 4
Drug: 5fluorouracil — Administered in accordance with local guidelines , prescribing information/summary of product
  Arms: Phase 1b: Dose Expansion: Cohort 6; Phase 1b: Dose Expansion: Cohort 7; Phase 1b: Dose Expansion: Cohort 9
Drug: Oxaliplatin — Administered in accordance with local guidelines , prescribing information/summary of product
  Arms: Phase 1b: Dose Expansion: Cohort 9
Drug: Capecitabine — Administered in accordance with local guidelines , prescribing information/summary of product
  Arms: Phase 1b: Dose Expansion: Cohort 9

SUMMARY:
The primary objectives of this study were: to assess the safety and tolerability, to determine the maximum tolerated dose (MTD) or maximum administered dose (MAD) and to determine the recommended Phase 2 dose (RP2D) of BGB-A1217 (known as ociperlimab) in combination with tislelizumab in participants with advanced solid tumors in phase 1.

Primary objective of Phase 1b was to assess overall response rate (ORR) determined by Investigator per Response Evaluation Criteria in Solid Tumors (RECIST) version (v).1.1 for patients in each dose-expansion cohort.

ELIGIBILITY:
Key Inclusion Criteria:

Phase 1 Key Inclusion Criteria

1. Had Eastern Cooperative Oncology Group (ECOG) Performance Status less than or equal to (<=) 1.
2. Greater than or equal to (>=) measurable lesion per RECIST v1.1.
3. Had adequate organ function.
4. Phase 1- Participants with histologically or cytologically confirmed advanced, metastatic, unresectable solid tumors who had previously received standard systemic therapy or for which treatment is not available, not tolerated or refused.

Phase 1b Key Inclusion Criteria

1. Signed informed consent form (ICF) and able to comply with study requirements.
2. Age >= 18 years (or the legal age of consent) at the time the ICF was signed.
3. Histologically or cytologically confirmed tumor types in the following disease cohorts:

   Cohort 1: stage IV squamous NSCLC Cohort 2: stage IV non-squamous NSCLC Cohort 3: stage IV squamous or non-squamous NSCLC with PD-L1 positive. Cohort 4: extensive-stage SCLC Cohort 5: stage IIIB, IIIC or IV NSCLC Cohort 6: stage IV ESCC Cohort 7: stage IV EAC Cohort 8: recurrent or metastatic HNSCC incurable by local therapies Cohort 9: stage IV G/GEJ adenocarcinoma. Cohort 10: stage IV squamous or non-squamous NSCLC with PD-L1 positive.
4. ECOG Performance Status <= 1
5. Adequate organ function
6. Were willing to use highly effective method of birth control

Phase 1 Key Exclusion Criteria:

1. Active brain or leptomeningeal metastasis.
2. Active autoimmune diseases or history of autoimmune diseases that could have relapsed.
3. Had severe chronic or active infections requiring systemic antibacterial, antifungal or antiviral therapy, including tuberculosis infection, etc. (antiviral therapy is permitted for patients with hepatocellular carcinoma).
4. Concurrent participation in another therapeutic clinical trial.
5. Received prior therapies targeting TIGIT.

Phase 1b Key Exclusion Criteria:

1. Participants with any prior therapy for recurrent/metastatic disease.
2. Non-squamous NSCLC patients with sensitizing epidermal growth factor receptor (EGFR) mutation, anaplastic lymphoma kinase (ALK) fusion, and c-ros oncogene 1 (ROS1) fusion.
3. Gastric cancer participants with squamous or with positive HER2 expression.
4. Prior therapy with any drug specifically targeting T-cell co-stimulation or checkpoint pathways. (anti-PD(L)1 exception for Cohort 5).
5. Active leptomeningeal disease or uncontrolled brain metastasis.
6. Active autoimmune diseases or history of autoimmune diseases that may relapse.
7. With severe chronic or active infections requiring systemic antibacterial, antifungal or antiviral therapy, including tuberculosis infection, etc. (antiviral therapy is permitted for participants with hepatocellular carcinoma).
8. Concurrent participation in another therapeutic clinical study.

NOTE: Other protocol-defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2024-08-07 (Actual); Study Completion 2024-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (65):
- United States (11):
  - Mayo Clinic Phoenix, Phoenix, Arizona
  - Scri Florida Cancer Specialists South, Fort Myers, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Scri Florida Cancer Specialists North, St. Petersburg, Florida
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Providence Portland Medical Center, Portland, Oregon
  - Tennessee Oncology, Pllc Nashville, Nashville, Tennessee
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (12):
  - Blacktown Cancer and Haematology Centre, Blacktown, New South Wales
  - Chris Obrien Lifehouse, Camperdown, New South Wales
  - Pindara Private Hospital, Benowa, Queensland
  - Icon Cancer Foundation, South Brisbane, Queensland
  - Metro South Health, Cancer Trials Unit Division of Cancer Services Pah, Woolloongabba, Queensland
  - Ashford Cancer Centre Research Northeast, Windsor Gardens, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Bendigo Health, Bendigo, Victoria
  - Monash Health, Clayton, Victoria
  - St Vincents Hospital, Fitzroy, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
  - St John of God Health Care, Subiaco, Western Australia
- China (23):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Tongren Hospital, Cmu, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Luhe Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi
  - Jinan Central Hospital, Jinan, Shandong
  - Weifang Peoples Hospital, Weifang, Shandong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital and Institute, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Nzcr Christchurch, Christchurch
- South Korea (8):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - The Catholic University of Korea, St Vincents Hospital, Suwon, Gyeonggi-do
  - Gyeongsang National University Hospital, Jinju, Gyeongsangnam-do
  - Gachon University Gil Medical Center, Incheon, Incheon Gwang'yeogsi
  - Severance Hospital Yonsei University Health System, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St Marys Hospital, Seoul, Seoul Teugbyeolsi
  - Smg Snu Boramae Medical Center, Seoul, Seoul Teugbyeolsi
- Taiwan (9):
  - Hualien Tzu Chi Hospital, Hualien City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - Veterans General Hospital Taichung, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Taipei Tzu Chi Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/

REFERENCES:
- [Result] Frentzas S, Kao S, Gao R, Zheng H, Rizwan A, Budha N, de la Hoz Pedroza L, Tan W, Meniawy T. AdvanTIG-105: a phase I dose escalation study of the anti-TIGIT monoclonal antibody ociperlimab in combination with tislelizumab in patients with advanced solid tumors. J Immunother Cancer. 2023 Oct;11(10):e005829. doi: 10.1136/jitc-2022-005829. PMID 37857528

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: Dose Escalation: Ociperlimab 50 mg + Tislelizumab 200 mg: Participants received ociperlimab 50 milligrams (mg) intravenous (IV) infusion on Day 1 of each cycle (cycle 1= 28 days) and tislelizumab 200 mg IV infusion on Day 8 of Cycle 1. If tolerated, participants received ociperlimab and tislelizumab doses IV on Cycle 2 Day 1 (cycle 2 onwards = 21 days) and thereafter every 21 days (that is, [i.e.], every 3 weeks [Q3W]) until disease progression, intolerable toxicity, or withdrawal of consent.
- Phase 1: Dose Escalation: Ociperlimab 900 mg + Tislelizumab 200 mg: Participants received ociperlimab 900 mg IV infusion on Day 1 of each cycle (cycle 1= 28 days) and tislelizumab 200 mg IV infusion on Day 8 of Cycle 1. If tolerated, participants received ociperlimab and tislelizumab doses IV on Cycle 2 Day 1 (cycle 2 onwards = 21 days) and thereafter every 21 days (i.e. Q3W) until disease progression, intolerable toxicity, or withdrawal of consent.
- Phase 1: Dose Verification: Cohort 1A (Ociperlimab 900 mg): Participants received ociperlimab 900 mg as monotherapy IV infusion on Day 1 of each 21-day treatment cycle until disease progression, intolerable toxicity, or withdrawal of consent.
- Phase 1: Dose Verification: Cohort 1B (Ociperlimab 900 mg + Tislelizumab 200 mg): Participants received ociperlimab 900 mg IV infusion on Day 1 of each 21-day treatment cycle and tislelizumab 200 mg IV infusion once every 21 days (i.e. Q3W) until disease progression, intolerable toxicity, or withdrawal of consent.
- Phase 1b: Dose Expansion: Cohort 1: Participants with metastatic squamous non-small cell lung cancer (NSCLC) received treatment with ociperlimab 900 mg IV infusion along with tislelizumab 200 mg IV infusion on Day 1 of each 21-day cycle. Participants also received 4 to 6 cycles of chemotherapy with carboplatin area under the curve (AUC) 5 or 6 (Day 1) + paclitaxel 200 or 175 mg/m^2 (Day 1) or nab paclitaxel 100 mg/m^2 (Days 1, 8 and 15) Q3W until disease progression, intolerable toxicity, or withdrawal of consent.
- Phase 1b: Dose Expansion: Cohort 2: Participants with metastatic non-squamous NSCLC received treatment with ociperlimab 900 mg IV infusion and tislelizumab 200 mg IV infusion on Day 1 of each 21-day cycle. Participants also received cisplatin 75 mg/m^2 or carboplatin (AUC 5) and pemetrexed 500 mg/m^2 (on Day 1) Q3W for 4-6 cycles followed by ociperlimab 900 mg + tislelizumab 200 mg + pemetrexed 500 mg/m^2 on Day 1 Q3W and were followed up until disease progression, intolerable toxicity, or withdrawal of consent.
- Phase 1b: Dose Expansion: Cohort 3: Participants with metastatic NSCLC (programmed cell death protein-ligand 1 [PD-L1] positive, tumour cells [TC] >=1%) were treated with ociperlimab 900 mg IV infusion and tislelizumab 200 mg IV infusion on Day 1 of each 21-day cycle until disease progression, intolerable toxicity, or withdrawal of consent.
- Phase 1b: Dose Expansion: Cohort 4: Participants with extensive-stage small-cell lung cancer (SCLC) received treatment with ociperlimab 900 mg IV infusion, tislelizumab 200 mg IV infusion. Participants also received 4 cycles of etoposide 100 mg/m^2 (on Days 1, 2, 3), and cisplatin 75 mg/m^2 /carboplatin AUC 5 (Day 1) Q3W, followed by ociperlimab 900 mg (Day 1) + tislelizumab 200 mg (Day 1) Q3W until disease progression, intolerable toxicity, or withdrawal of consent.
- Phase 1b: Dose Expansion: Cohort 5: Checkpoint inhibitor (CPI)-experienced NSCLC participants received treatment with ociperlimab 900 mg IV infusion and tislelizumab 200 mg IV infusions on Day 1 of each 21-day cycle until disease progression, intolerable toxicity, or withdrawal of consent.
- Phase 1b: Dose Expansion: Cohort 6: Participants with metastatic esophageal squamous cell carcinoma (ESCC) received treatment with 6 cycles of ociperlimab 900 mg (Day 1) IV infusion, tislelizumab 200 mg (Day 1) IV infusion, cisplatin 75 mg/m^2 (Day 1), and Fluorouracil 750-800 mg/m^2 (5-FU; Day 1 to Day 5) or paclitaxel 200 or 175 mg/m^2 (Day 1) Q3W followed by ociperlimab 900 mg and tislelizumab 200 mg on Day 1 of every 21-day cycle until disease progression, intolerable toxicity, or withdrawal of consent.
- Phase 1b: Dose Expansion: Cohort 7: Participants with metastatic esophageal adenocarcinoma (EAC) received treatment with 6 cycles of ociperlimab 900 mg (Day 1) IV infusion, tislelizumab 200 mg (Day 1) IV infusion, cisplatin 75 mg/m^2 (Day 1), and Fluorouracil 750-800 mg/m^2 (5-FU; Day 1 to Day 5) or paclitaxel 200 or 175 mg/m^2 (Day 1) Q3W followed by ociperlimab 900 mg and tislelizumab 200 mg on Day 1 of every 21-day cycle until disease progression, intolerable toxicity, or withdrawal of consent.
- Phase 1b: Dose Expansion: Cohort 8: Participants with recurrent or metastatic head and neck squamous cell carcinoma (HNSCC; PD-L1 positive, visually estimated Combined Positive Score [vCPS] >= 1%) received treatment with ociperlimab 900 mg IV infusion and tislelizumab 200 mg IV infusions on Day 1 of every 21-day cycle until disease progression, intolerable toxicity, or withdrawal of consent.
- Phase 1b: Dose Expansion: Cohort 9: Participants with unresectable, locally advanced, recurrent, or metastatic gastric or gastroesophageal junction (G/GEJ) adenocarcinoma received treatment with 6 cycles of ociperlimab 900 mg (Day 1) IV infusion, tislelizumab 200 mg (Day 1) IV infusion, (oxaliplatin 1300 mg/m^2 [Day 1] and capecitabine 1000 mg/m^2 [Day 1-14 twice daily], or cisplatin 75 mg/m^2 [Day], and 5-FU 750-800 mg/m^2 [Day 1-5]) Q3W followed by ociperlimab 900 mg (Day 1), tislelizumab 200 mg (Day 1) + capecitabine 1000 mg/m^2 twice daily (Day 1-14) Q3W until disease progression, intolerable toxicity, or withdrawal of consent.
- Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 450 mg + Tislelizumab 200 mg): Participants with metastatic NSCLC (PD-L1 positive, TC >= 1%) received treatment with ociperlimab 450 mg IV infusion and tislelizumab 200 mg IV infusion on Day 1 of every 21-day cycle until disease progression, intolerable toxicity, or withdrawal of consent.
- Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 900 mg + Tislelizumab 200 mg): Participants with metastatic NSCLC (PD-L1 positive, TC >= 1%) received treatment with ociperlimab 900 mg IV infusion and tislelizumab 200 mg IV infusion on Day 1 of every 21-day cycle until disease progression, intolerable toxicity, or withdrawal of consent.
- Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 1800 mg + Tislelizumab 200 mg): Participants with metastatic NSCLC (PD-L1 positive, TC >= 1%) received treatment with ociperlimab 1800 mg IV infusion and tislelizumab 200 mg IV infusion on Day 1 of every 21-day cycle until disease progression, intolerable toxicity, or withdrawal of consent.
Period: Overall Study
Arm/Group | Phase 1: Dose Escalation: Ociperlimab 50 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 150 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 450 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 900 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 1800 mg + Tislelizumab 200 mg | Phase 1: Dose Verification: Cohort 1A (Ociperlimab 900 mg) | Phase 1: Dose Verification: Cohort 1B (Ociperlimab 900 mg + Tislelizumab 200 mg) | Phase 1b: Dose Expansion: Cohort 1 | Phase 1b: Dose Expansion: Cohort 2 | Phase 1b: Dose Expansion: Cohort 3 | Phase 1b: Dose Expansion: Cohort 4 | Phase 1b: Dose Expansion: Cohort 5 | Phase 1b: Dose Expansion: Cohort 6 | Phase 1b: Dose Expansion: Cohort 7 | Phase 1b: Dose Expansion: Cohort 8 | Phase 1b: Dose Expansion: Cohort 9 | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 450 mg + Tislelizumab 200 mg) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 900 mg + Tislelizumab 200 mg) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 1800 mg + Tislelizumab 200 mg)
Started | 1 | 3 | 6 | 16 | 6 | 9 | 11 | 41 | 43 | 45 | 43 | 26 | 21 | 6 | 41 | 60 | 24 | 21 | 23
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 3 | 6 | 16 | 6 | 9 | 11 | 41 | 43 | 45 | 43 | 26 | 21 | 6 | 41 | 60 | 24 | 21 | 23
Not completed — Death | 0 | 0 | 4 | 7 | 2 | 4 | 3 | 24 | 24 | 22 | 35 | 18 | 14 | 6 | 19 | 42 | 9 | 8 | 10
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 5 | 2 | 0 | 1 | 0 | 4 | 4 | 4 | 2 | 3 | 0 | 9 | 5 | 1 | 3 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 0 | 2 | 2 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Completed all Assessments | 1 | 3 | 1 | 3 | 2 | 5 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 10 | 18 | 3 | 3 | 4 | 0 | 7 | 8 | 9 | 7 | 8
Not completed — Transfer to a Company Sponsored Clinical Trial | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 5 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 2
Not completed — Transfer to Patient Supply Treatment Program (PTS) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis included participants from safety analysis set, that is, (i.e.) participants who received more than or equal to (>=) 1 dose of any study drug.
Groups:
- Phase 1: Dose Escalation: Ociperlimab 50 mg + Tislelizumab 200 mg: Participants received ociperlimab 50 mg IV infusion on Day 1 of each cycle (cycle 1= 28 days) and tislelizumab 200 mg IV infusion on Day 8 of Cycle 1. If tolerated, participants received ociperlimab and tislelizumab doses IV on Cycle 2 Day 1 (cycle 2 onwards = 21 days) and thereafter every 21 days (i.e., Q3W) until disease progression, intolerable toxicity, or withdrawal of consent.
- Phase 1b: Dose Expansion: Cohort 1: Participants with metastatic squamous NSCLC received treatment with ociperlimab 900 mg IV infusion along with tislelizumab 200 mg IV infusion on Day 1 of each 21-day cycle. Participants also received 4 to 6 cycles of chemo with carboplatin AUC 5 or 6 (Day 1) + paclitaxel 200 or 175 mg/m^2 (Day 1) or nab paclitaxel 100 mg/m^2 (Days 1, 8 and 15) Q3W until disease progression, intolerable toxicity, or withdrawal of consent.
- Phase 1b: Dose Expansion: Cohort 2: Participants with metastatic non-squamous NSCLC received treatment with ociperlimab 900 mg IV infusion and tislelizumab 200 mg IV infusion on Day 1 of each 21-day cycle. Participants also received cisplatin 75 mg/m^2 or carboplatin (AUC 5) and pemetrexed 500 mg/m^2 (on Day 1) Q3W for 4-6 cycles followed by ociperlimab 900 mg + tislelizumab 200 mg + pemetrexed 500 mg/m^2 on Day 1 Q3W until disease progression, intolerable toxicity, or withdrawal of consent.
- Phase 1b: Dose Expansion: Cohort 3: Participants with metastatic NSCLC (PD-L1 positive, TC >=1%) were treated with ociperlimab 900 mg IV infusion and tislelizumab 200 mg IV infusion on Day 1 of each 21-day cycle until disease progression, intolerable toxicity, or withdrawal of consent.
- Phase 1b: Dose Expansion: Cohort 4: Participants with extensive-stage SCLC received treatment with ociperlimab 900 mg IV infusion, tislelizumab 200 mg IV infusion. Participants also received 4 cycles of etoposide 100 mg/m^2 (on Days 1, 2, 3), and cisplatin 75 mg/m^2 /carboplatin AUC 5 (Day 1) Q3W, followed by ociperlimab 900 mg (Day 1) + tislelizumab 200 mg (Day 1) Q3W until disease progression, intolerable toxicity, or withdrawal of consent.
- Phase 1b: Dose Expansion: Cohort 6: Participants with metastatic ESCC received treatment with 6 cycles of ociperlimab 900 mg (Day 1) IV infusion, tislelizumab 200 mg (Day 1) IV infusion, cisplatin 75 mg/m^2 (Day 1), and Fluorouracil 750-800 mg/m^2 (5-FU; Day 1 to Day 5) or paclitaxel 200 or 175 mg/m^2 (Day 1) Q3W followed by ociperlimab 900 mg and tislelizumab 200 mg on Day 1 of every 21-day cycle and were followed up until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
- Phase 1b: Dose Expansion: Cohort 7: Participants with metastatic EAC received treatment with 6 cycles of ociperlimab 900 mg (Day 1) IV infusion, tislelizumab 200 mg (Day 1) IV infusion, cisplatin 75 mg/m^2 (Day 1), and Fluorouracil 750-800 mg/m^2 (5-FU; Day 1 to Day 5) or paclitaxel 200 or 175 mg/m^2 (Day 1) Q3W followed by ociperlimab 900 mg and tislelizumab 200 mg on Day 1 of every 21-day cycle until disease progression, intolerable toxicity, or withdrawal of consent.
- Phase 1b: Dose Expansion: Cohort 8: Participants with recurrent or metastatic HNSCC; PD-L1 positive, vCPS >= 1%) received treatment with ociperlimab 900 mg IV infusion and tislelizumab 200 mg IV infusions on Day 1 of every 21-day cycle until disease progression, intolerable toxicity, or withdrawal of consent.
- Phase 1b: Dose Expansion: Cohort 9: Participants with unresectable, locally advanced, recurrent, or metastatic G/GEJ adenocarcinoma received treatment with 6 cycles of ociperlimab 900 mg (Day 1) IV infusion, tislelizumab 200 mg (Day 1) IV infusion, (oxaliplatin 1300 mg/m^2 [Day 1] and capecitabine 1000 mg/m^2 [Day 1-14 twice daily], or cisplatin 75 mg/m^2 [Day 1], and 5-FU 750-800 mg/m^2 [Day 1-5]) Q3W followed by ociperlimab 900 mg (Day 1), tislelizumab 200 mg (Day 1) + capecitabine 1000 mg/m^2 twice daily (Day 1-14) Q3W until disease progression, intolerable toxicity, or withdrawal of consent.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Dose Escalation: Ociperlimab 50 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 150 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 450 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 900 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 1800 mg + Tislelizumab 200 mg | Phase 1: Dose Verification: Cohort 1A (Ociperlimab 900 mg) | Phase 1: Dose Verification: Cohort 1B (Ociperlimab 900 mg + Tislelizumab 200 mg) | Phase 1b: Dose Expansion: Cohort 1 | Phase 1b: Dose Expansion: Cohort 2 | Phase 1b: Dose Expansion: Cohort 3 | Phase 1b: Dose Expansion: Cohort 4 | Phase 1b: Dose Expansion: Cohort 5 | Phase 1b: Dose Expansion: Cohort 6 | Phase 1b: Dose Expansion: Cohort 7 | Phase 1b: Dose Expansion: Cohort 8 | Phase 1b: Dose Expansion: Cohort 9 | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 450 mg + Tislelizumab 200 mg) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 900 mg + Tislelizumab 200 mg) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 1800 mg + Tislelizumab 200 mg) | Total
Number analyzed (Participants) | 1 | 3 | 6 | 16 | 6 | 9 | 11 | 41 | 43 | 45 | 43 | 26 | 21 | 6 | 41 | 60 | 24 | 21 | 23 | 446
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (NA) — Standard deviation could not be calculated as only one participant was available for analysis. | 48.7 (18.90) | 56.8 (11.25) | 53.3 (14.75) | 67.0 (6.90) | 61.9 (7.66) | 60.4 (11.45) | 64.9 (8.04) | 62.7 (8.71) | 65.4 (8.59) | 63.6 (9.79) | 66.7 (9.34) | 62.2 (6.02) | 63.0 (4.24) | 63.5 (10.74) | 60.1 (11.65) | 61.5 (10.46) | 64.0 (7.05) | 65.4 (8.98) | 62.8 (10.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 4 | 10 | 2 | 3 | 1 | 6 | 12 | 16 | 11 | 8 | 3 | 0 | 6 | 16 | 7 | 4 | 6 | 116
  Male | 1 | 2 | 2 | 6 | 4 | 6 | 10 | 35 | 31 | 29 | 32 | 18 | 18 | 6 | 35 | 44 | 17 | 17 | 17 | 330
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 4
  Not Hispanic or Latino | 1 | 3 | 6 | 16 | 6 | 9 | 11 | 41 | 43 | 44 | 43 | 26 | 21 | 6 | 41 | 58 | 24 | 20 | 22 | 441
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 2 | 3 | 1 | 9 | 11 | 38 | 35 | 34 | 32 | 11 | 16 | 0 | 37 | 46 | 22 | 19 | 17 | 333
  Native Hawaiian or other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 1 | 2 | 4 | 13 | 4 | 0 | 0 | 2 | 7 | 9 | 8 | 15 | 2 | 6 | 2 | 11 | 1 | 2 | 6 | 95
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
  Not Reported/Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 4
  Multiple | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 9
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An AE was defined as any unfavorable and unintended sign, symptom, or disease associated with the use of study drugs, whether considered related to study drugs or not. A serious adverse event (SAE) was any untoward medical occurrence that, at any dose, resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability, was a congenital anomaly or was considered a medically significant. Treatment-emergent adverse event (TEAE) was an AE that has an onset date or a worsening in severity from baseline on or after the first dose of study drug up to 30 days following study drug discontinuation or initiation of the first new systemic anticancer therapy, whichever occurred first. Severity of AEs was assessed according to National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI-CTCAE) v.5.0, which consists of: Grade 1 Mild; Grade 2 Moderate; Grade 3: Severe; Grade 4: Life-threatening; Grade 5: Death due to AE.
Time Frame: Up to 30 days after the last dose of study interventions (up to 35.7 months [Dose escalation cohorts] and up to 13.3 months [Dose verification cohorts])
Population: Analysis was performed on the safety analysis set that included all participants who received >= 1 dose of any study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: Dose Escalation: Ociperlimab 50 mg + Tislelizumab 200 mg: Participants received ociperlimab 50 mg IV infusion on Day 1 of each cycle (cycle 1= 28 days) and tislelizumab 200 mg IV infusion on Day 8 of Cycle 1. If tolerated, participants received ociperlimab and tislelizumab IV on Cycle 2 Day 1 (cycle 2 onwards = 21 days) and thereafter every 21 days (i.e., Q3W) until disease progression, intolerable toxicity, or withdrawal of consent.
Arm/Group | Phase 1: Dose Escalation: Ociperlimab 50 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 150 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 450 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 900 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 1800 mg + Tislelizumab 200 mg | Phase 1: Dose Verification: Cohort 1A (Ociperlimab 900 mg) | Phase 1: Dose Verification: Cohort 1B (Ociperlimab 900 mg + Tislelizumab 200 mg)
Number analyzed (Participants) | 1 | 3 | 6 | 16 | 6 | 9 | 11
Participants
  Participants with any TEAE | 1 | 3 | 6 | 15 | 6 | 9 | 11
  Participants with >= Grade 3 TEAE | 1 | 2 | 4 | 11 | 2 | 4 | 5
  Serious TEAE | 1 | 2 | 3 | 9 | 1 | 3 | 5

2. Primary Outcome: Phase 1: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: The DLTs were defined as high grade (Grade 3 or 4) non-hematologic toxicities (that is, >= Grade 4 toxicity; Grade 3 toxicity that is clinically significant and does not resolve to baseline or <=Grade 1 within 7 days of initiating optimal supportive care), or hematologic toxicities (Grade 4 neutropenia lasting > 7 days; >=Grade 3 febrile neutropenia; Grade 3 thrombocytopenia with clinically significant bleeding; Grade 4 thrombocytopenia lasting > 7 days; >=Grade 4 anemia occurring during the DLT assessment window and considered by the investigator to be related to ociperlimab and/or tislelizumab.
Time Frame: Up to 28 days (for Dose escalation cohorts) and up to 21 days (for Dose verification cohorts)
Population: Analysis was performed on the safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Dose Escalation: Ociperlimab 50 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 150 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 450 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 900 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 1800 mg + Tislelizumab 200 mg | Phase 1: Dose Verification: Cohort 1A (Ociperlimab 900 mg) | Phase 1: Dose Verification: Cohort 1B (Ociperlimab 900 mg + Tislelizumab 200 mg)
Number analyzed (Participants) | 1 | 3 | 6 | 16 | 6 | 9 | 11
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Phase 1: Maximum Administered Dose (MAD) of Ociperlimab in Combination With Tislelizumab
Description: MAD was defined as the highest dose of ociperlimab administered.
Time Frame: Up to 28 days (Dose escalation cohort)
Population: Analysis was performed on the safety analysis set.
Measure: Number; unit: milligram (mg)
Groups:
- Phase 1: Dose Escalation: All Participants: All participants who received ociperlimab escalated doses (50,150, 450, 900 and 1800 mg) through IV infusion on Day 1 of each cycle (cycle 1= 28 days) and tislelizumab 200 mg IV infusion on Day 8 of Cycle 1. If tolerated, participants received ociperlimab and tislelizumab doses IV on Cycle 2 Day 1 (cycle 2 onwards = 21 days) and thereafter every 21 days (i.e., Q3W) until disease progression, intolerable toxicity, or withdrawal of consent.
Arm/Group | Phase 1: Dose Escalation: All Participants
Number analyzed (Participants) | 32
milligram (mg) | 1800

4. Primary Outcome: Phase 1: Recommended Phase 2 Dose (RP2D) of Ociperlimab in Combination With Tislelizumab
Description: RP2D of Ociperlimab in combination with Tislelizumab 200 mg was determined primarily from the safety, tolerability, and pharmacokinetic (PK) data of dose escalation cohorts.
Time Frame: up to 28 days (Dose escalation cohorts)
Population: Analysis was performed on the safety analysis set.
Measure: Number; unit: mg
Arm/Group | Phase 1: Dose Escalation: All Participants
Number analyzed (Participants) | 32
mg | 900

5. Primary Outcome: Phase 1b: Overall Response Rate (ORR) as Per Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1
Description: ORR was defined as the percentage of participants who had complete response (CR) or partial response (PR). Per Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1., CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Maximum time duration on study: up to 41.6 months (Cohorts 1 to 9) and up to 21.4 months (Cohort 10)
Population: Analysis was performed on efficacy evaluable analysis set that included all treated participants who had measurable disease at baseline and >= 1 evaluable postbaseline tumor response assessment unless discontinued from any component of study treatment due to clinical progression of disease (PD) or death within 7 weeks after first dose.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase 1b: Dose Expansion: Cohort 5: CPI-experienced NSCLC participants received treatment with ociperlimab 900 mg IV infusion and tislelizumab 200 mg IV infusions on Day 1 of each 21-day cycle until disease progression, intolerable toxicity, or withdrawal of consent.
- Phase 1b: Dose Expansion: Cohort 6: Participants with metastatic ESCC received treatment with 6 cycles of ociperlimab 900 mg (Day 1) IV infusion, tislelizumab 200 mg (Day 1) IV infusion, cisplatin 75 mg/m^2 (Day 1), and Fluorouracil 750-800 mg/m^2 (5-FU; Day 1 to Day 5) or paclitaxel 200 or 175 mg/m^2 (Day 1) Q3W followed by ociperlimab 900 mg and tislelizumab 200 mg on Day 1 of every 21-day cycle until disease progression, intolerable toxicity, or withdrawal of consent.
- Phase 1b: Dose Expansion: Cohort 8: Participants with recurrent or metastatic HNSCC (PD-L1 positive, vCPS >= 1%) received treatment with ociperlimab 900 mg IV infusion and tislelizumab 200 mg IV infusions on Day 1 of every 21-day cycle until disease progression, intolerable toxicity, or withdrawal of consent.
- Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 450 mg + Tislelizumab 200 mg): Participants with metastatic NSCLC (PD-L1 positive, TC >= 1%) received treatment with ociperlimab 450 mg IV infusion and tislelizumab 200 mg IV infusion on Day 1 of every 21-day cycle and were followed up until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
- Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 900 mg + Tislelizumab 200 mg): Participants with metastatic NSCLC (PD-L1 positive, TC >= 1%) received treatment with ociperlimab 900 mg IV infusion and tislelizumab 200 mg IV infusion on Day 1 of every 21-day cycle and were followed up until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
Arm/Group | Phase 1b: Dose Expansion: Cohort 1 | Phase 1b: Dose Expansion: Cohort 2 | Phase 1b: Dose Expansion: Cohort 3 | Phase 1b: Dose Expansion: Cohort 4 | Phase 1b: Dose Expansion: Cohort 5 | Phase 1b: Dose Expansion: Cohort 6 | Phase 1b: Dose Expansion: Cohort 7 | Phase 1b: Dose Expansion: Cohort 8 | Phase 1b: Dose Expansion: Cohort 9 | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 450 mg + Tislelizumab 200 mg) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 900 mg + Tislelizumab 200 mg) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 1800 mg + Tislelizumab 200 mg)
Number analyzed (Participants) | 40 | 42 | 45 | 41 | 26 | 19 | 6 | 39 | 59 | 23 | 19 | 23
percentage of participants | 55 [38.5 to 70.7] | 54.8 [38.7 to 70.2] | 40.0 [25.7 to 55.7] | 65.9 [49.4 to 79.9] | 7.7 [0.9 to 25.1] | 68.4 [43.4 to 87.4] | 33.3 [4.3 to 77.7] | 33.3 [19.1 to 50.2] | 50.8 [37.5 to 64.1] | 34.8 [16.4 to 57.3] | 26.3 [9.1 to 51.2] | 34.8 [16.4 to 57.3]

6. Secondary Outcome: Phase 1: ORR as Per RECIST v.1.1
Description: ORR was defined as the percentage of participants who had CR or PR as determined from investigator-derived tumor assessments per RECIST v. 1.1. Per RECIST v.1.1., CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Maximum time duration on study: up to 35.7 months (Dose escalation cohorts) and up to 13.3 months (Dose verification cohorts)
Population: Analysis was performed on efficacy evaluable analysis set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: Dose Escalation: Ociperlimab 50 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 150 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 450 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 900 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 1800 mg + Tislelizumab 200 mg | Phase 1: Dose Verification: Cohort 1A (Ociperlimab 900 mg) | Phase 1: Dose Verification: Cohort 1B (Ociperlimab 900 mg + Tislelizumab 200 mg)
Number analyzed (Participants) | 1 | 3 | 6 | 16 | 5 | 9 | 10
percentage of participants | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 70.8] | 16.7 [0.4 to 64.1] | 6.3 [0.2 to 30.2] | 20 [0.5 to 71.6] | 0.0 [0.0 to 33.6] | 10 [0.3 to 44.5]

7. Secondary Outcome: Phase 1: Duration of Response (DOR) as Per RECIST v.1.1
Description: DOR was defined as the time from the first determination of an overall response per RECIST v1.1 until the first documentation of progression (PD) or death, whichever came first. DOR was estimated using the Kaplan-Meier method. Per RECIST v.1.1., CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study.
Time Frame: From the first determination of an overall response until PD or death, whichever came first (Maximum time duration on study: up to 35.7 months [Dose escalation cohorts] and up to 13.3 months [Dose verification cohorts])
Population: Analysis was performed on participants in the efficacy evaluable analysis set with an objective response. Here, "0" in the overall number of participants analyzed signifies no participants with available data at the specified time-points.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1: Dose Escalation: Ociperlimab 50 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 150 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 450 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 900 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 1800 mg + Tislelizumab 200 mg | Phase 1: Dose Verification: Cohort 1A (Ociperlimab 900 mg) | Phase 1: Dose Verification: Cohort 1B (Ociperlimab 900 mg + Tislelizumab 200 mg)
Number analyzed (Participants) | 0 | 0 | 1 | 1 | 1 | 0 | 1
months |  |  | 2.8 [NA to NA] — 95% Confidence Interval (CI) could not be calculated due to an insufficient number of participants with events. | 3.6 [NA to NA] — 95% CI could not be calculated due to an insufficient number of participants with events. | 8.4 [NA to NA] — 95% CI could not be calculated due to an insufficient number of participants with events. |  | 7 [NA to NA] — 95% CI could not be calculated due to an insufficient number of participants with events.

8. Secondary Outcome: Phase 1: Disease Control Rate (DCR) as Per RECIST v.1.1
Description: DCR was defined as the percentage of participants with best overall response (BOR), as per RECIST v.1.1, of a CR, PR, or stable disease (SD). Per RECIST v.1.1., CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: as for outcome 7
Population: Analysis was performed on efficacy evaluable analysis set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase 1: Dose Escalation: Ociperlimab 150 mg + Tislelizumab 200 mg: Participants received ociperlimab 150 mg IV infusion on Day 1 of each cycle (cycle 1= 28 days) and tislelizumab 200 mg IV infusion on Day 8 of Cycle 1. If tolerated, participants received ociperlimab and tislelizumab IV on Cycle 2 Day 1 (cycle 2 onwards = 21 days) and thereafter every 21 days (i.e. Q3W) until disease progression, intolerable toxicity, or withdrawal of consent.
- Phase 1: Dose Escalation: Ociperlimab 450 mg + Tislelizumab 200 mg: Participants received ociperlimab 450 mg IV infusion on Day 1 of each cycle (cycle 1= 28 days) and tislelizumab 200 mg IV infusion on Day 8 of Cycle 1. If tolerated, participants received ociperlimab and tislelizumab IV on Cycle 2 Day 1 (cycle 2 onwards = 21 days) and thereafter every 21 days (i.e. Q3W) until disease progression, intolerable toxicity, or withdrawal of consent.
- Phase 1: Dose Escalation: Ociperlimab 900 mg + Tislelizumab 200 mg: Participants received ociperlimab 900 mg IV infusion on Day 1 of each cycle (cycle 1= 28 days) and tislelizumab 200 mg IV infusion on Day 8 of Cycle 1. If tolerated, participants received ociperlimab and tislelizumab IV on Cycle 2 Day 1 (cycle 2 onwards = 21 days) and thereafter every 21 days (i.e. Q3W) until disease progression, intolerable toxicity, or withdrawal of consent.
- Phase 1: Dose Escalation: Ociperlimab 1800 mg + Tislelizumab 200 mg: Participants received ociperlimab 1800 mg IV infusion on Day 1 of each cycle (cycle 1= 28 days) and tislelizumab 200 mg IV infusion on Day 8 of Cycle 1. If tolerated, participants received ociperlimab and tislelizumab IV on Cycle 2 Day 1 (cycle 2 onwards = 21 days) and thereafter every 21 days (i.e. Q3W) until disease progression, intolerable toxicity, or withdrawal of consent.
Arm/Group | Phase 1: Dose Escalation: Ociperlimab 50 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 150 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 450 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 900 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 1800 mg + Tislelizumab 200 mg | Phase 1: Dose Verification: Cohort 1A (Ociperlimab 900 mg) | Phase 1: Dose Verification: Cohort 1B (Ociperlimab 900 mg + Tislelizumab 200 mg)
Number analyzed (Participants) | 1 | 3 | 6 | 16 | 5 | 9 | 10
percentage of participants | 0 [0 to 97.5] | 33.3 [0.8 to 90.6] | 50 [11.8 to 88.2] | 50 [24.7 to 75.3] | 40 [5.3 to 85.3] | 33.3 [7.5 to 70.1] | 50 [18.7 to 81.3]

9. Secondary Outcome: Phase 1 (Dose Escalation): Serum Concentrations of Ociperlimab
Description: Serum concentrations of ociperlimab were measured. Post-dose refers to the data collected for 30 minutes post-infusion. "C" in the timeframe below refers to "Cycle" and D refers to "Day" and "h" refers to "hours".
Time Frame: C1D1 (pre and post dose; 24 hours (h) 72h, 168h and 336 h post-dose), C2D1 (pre- and post-dose), C5D1 (pre and post dose,168h and 336 h post-dose), C6D1 (pre and post-dose), pre-dose on C9D1,C13D1,C17D1,C25D1 (Cycle 1= 28 days; Cycle 2 onwards= 21 days)
Population: Analysis was performed on the pharmacokinetic (PK) analysis set that included all participants who received >= 1 dose of any component of study drugs per the protocol, and for whom any corresponding post-dose PK data were available. Here, number analyzed' = participants with available data of serum concentrations and "0" in the number analyzed signifies no participants with available data at specified time-points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Phase 1: Dose Escalation: Ociperlimab 50 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 150 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 450 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 900 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 1800 mg + Tislelizumab 200 mg
Number analyzed (Participants) | 1 | 3 | 6 | 16 | 6
micrograms per milliliter (mcg/mL)
  Cycle 1 Day 1- Pre-dose | NA (NA) — Geometric mean and Geometric coefficient of variation (GCV) could not be calculated due to an insufficient number of participants with lower limit of quantification (LLOQ) for analysis. | NA (NA) — Geometric mean and GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis. | NA (NA) — Geometric mean and GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis. | NA (NA) — Geometric mean and GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis. | NA (NA) — Geometric mean and GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis.
  Cycle 1 Day 1 post-dose: number analyzed (Participants) | 1 | 2 | 6 | 16 | 6
  Cycle 1 Day 1 post-dose | 14.70 (NA) — GCV could not be calculated due to an insufficient number of participants with events. | 44.59 (32) | 130.22 (19) | 259.66 (21) | 525.97 (29)
  Cycle 1 Day 1- 24 h | 10.30 (NA) — GCV could not be calculated due to an insufficient number of participants with events. | 31.67 (16) | 98.28 (16) | 198.72 (14) | 374.44 (29)
  Cycle 1 Day 1- 72 h | 6.49 (NA) — GCV could not be calculated due to an insufficient number of participants with events. | 18.43 (20) | 64.36 (29) | 136.15 (12) | 256.28 (35)
  Cycle 1 Day 1- 168 h: number analyzed (Participants) | 1 | 3 | 6 | 15 | 6
  Cycle 1 Day 1- 168 h | 2.58 (NA) — GCV could not be calculated due to an insufficient number of participants with events. | 11.49 (13) | 41.16 (43) | 90.08 (23) | 150.95 (31)
  Cycle 1 Day 1- 336 h: number analyzed (Participants) | 1 | 3 | 5 | 14 | 6
  Cycle 1 Day 1- 336 h | 1.34 (NA) — GCV could not be calculated due to an insufficient number of participants with events. | 7.03 (28) | 29.30 (46) | 64.72 (21) | 101.42 (40)
  Cycle 2 Day 1- Pre-dose: number analyzed (Participants) | 1 | 3 | 6 | 14 | 3
  Cycle 2 Day 1- Pre-dose | 0.33 (NA) — GCV could not be calculated due to an insufficient number of participants with events. | 2.23 (42) | 8.71 (109) | 24.96 (71) | 23.85 (87)
  Cycle 2 Day 1- Post-dose: number analyzed (Participants) | 1 | 3 | 6 | 14 | 3
  Cycle 2 Day 1- Post-dose | 13.90 (NA) — GCV could not be calculated due to an insufficient number of participants with events. | 48.11 (39) | 145.89 (30) | 277.69 (20) | 460.48 (45)
  Cycle 5 Day 1- Pre-dose: number analyzed (Participants) | 0 | 1 | 3 | 4 | 3
  Cycle 5 Day 1- Pre-dose |  | 5.44 (NA) — GCV could not be calculated due to an insufficient number of participants with events. | 28.39 (45) | 46.15 (108) | 121.94 (29)
  Cycle 5 Day 1- post-dose: number analyzed (Participants) | 0 | 1 | 2 | 4 | 3
  Cycle 5 Day 1- post-dose |  | 35.60 (NA) — GCV could not be calculated due to an insufficient number of participants with events. | 156.97 (3) | 298.93 (19) | 589.07 (19)
  Cycle 5 Day 1- 168 h: number analyzed (Participants) | 0 | 1 | 2 | 4 | 2
  Cycle 5 Day 1- 168 h |  | 15.30 (NA) — GCV could not be calculated due to an insufficient number of participants with events. | 77.59 (14) | 140.04 (35) | 265.52 (26)
  Cycle 5 Day 1- 336 h: number analyzed (Participants) | 0 | 1 | 2 | 4 | 2
  Cycle 5 Day 1- 336 h |  | 8.38 (NA) — GCV could not be calculated due to an insufficient number of participants with events. | 55.27 (8) | 96.09 (54) | 179.05 (36)
  Cycle 6 Day 1- Pre-dose: number analyzed (Participants) | 0 | 1 | 3 | 4 | 2
  Cycle 6 Day 1- Pre-dose |  | 6.94 (NA) — GCV could not be calculated due to an insufficient number of participants with events. | 23.92 (102) | 66.59 (64) | 154.07 (11)
  Cycle 6 Day 1- post-dose: number analyzed (Participants) | 0 | 1 | 3 | 4 | 2
  Cycle 6 Day 1- post-dose |  | 40.40 (NA) — GCV could not be calculated due to an insufficient number of participants with events. | 150.44 (19) | 343.48 (23) | 726.95 (8)
  Cycle 9 Day 1- Pre-dose: number analyzed (Participants) | 0 | 1 | 3 | 2 | 2
  Cycle 9 Day 1- Pre-dose |  | 7.57 (NA) — GCV could not be calculated due to an insufficient number of participants with events. | 36.98 (20) | 49.92 (41) | 140.64 (10)
  Cycle 13 Day 1- Pre-dose: number analyzed (Participants) | 0 | 1 | 1 | 1 | 2
  Cycle 13 Day 1- Pre-dose |  | 8.12 (NA) — GCV could not be calculated due to an insufficient number of participants with events. | 44.80 (NA) — GCV could not be calculated due to an insufficient number of participants with events. | 66.70 (NA) — GCV could not be calculated due to an insufficient number of participants with events. | 80.56 (111)
  Cycle 17 Day1- Pre-dose: number analyzed (Participants) | 0 | 0 | 1 | 0 | 2
  Cycle 17 Day1- Pre-dose |  |  | 45.50 (NA) — GCV could not be calculated due to an insufficient number of participants with events. |  | 113.00 (0.0000)
  Cycle 25 Day 1- Pre-dose: number analyzed (Participants) | 0 | 1 | 1 | 0 | 0
  Cycle 25 Day 1- Pre-dose |  | 9.05 (NA) — GCV could not be calculated due to an insufficient number of participants with events. | 47.20 (NA) — GCV could not be calculated due to an insufficient number of participants with events. |  |

10. Secondary Outcome: Phase 1 (Dose Escalation): Serum Concentrations of Tislelizumab
Description: Serum Concentrations of Tislelizumab was determined. Post-dose refers to the data collected for 30 minutes post-infusion.
Time Frame: Cycle 1, Day 8 (pre-dose), Cycle 1, Day 8 (post-dose), Cycle 2, Day 1 (pre-dose), Cycle 5 Day 1 (pre-dose), Cycle 5 Day 1 (post-dose), pre-dose of Cycle 6 Day 1, Cycle 9 Day 1, Cycle 13 Day 1, Cycle 17 Day 1, Cycle 25 Day 1 (each cycle = 21 days)
Population: Analysis was performed on PK analysis set. Here, number analyzed' = participants with available data for the analysis of serum concentrations and "0" in the number analyzed signifies no participant were available for analysis at specified time-points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Phase 1: Dose Escalation: Ociperlimab 50 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 150 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 450 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 900 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 1800 mg + Tislelizumab 200 mg
Number analyzed (Participants) | 1 | 3 | 6 | 16 | 6
micrograms per milliliter (mcg/mL)
  Cycle 1 Day 8 Predose: number analyzed (Participants) | 1 | 3 | 6 | 15 | 6
  Cycle 1 Day 8 Predose | 0.45 (NA) — GCV could not be calculated due to an insufficient number of participants available for analysis. | 16.50 (NA) — GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis. | 14.46 (350) | 18.60 (528) | NA (NA) — Geometric mean and GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis.
  Cycle 1 Day 8 Post-dose | 54.60 (NA) — GCV could not be calculated due to an insufficient number of participants available for analysis. | 62.89 (38) | 82.34 (48) | 67.93 (46) | 60.28 (27)
  Cycle 2 Day 1 Predose: number analyzed (Participants) | 1 | 3 | 6 | 14 | 3
  Cycle 2 Day 1 Predose | 11.50 (NA) — GCV could not be calculated due to an insufficient number of participants available for analysis. | 14.17 (69) | 20.05 (93) | 18.61 (82) | 10.37 (72)
  Cycle 5 Day 1 Predose: number analyzed (Participants) | 0 | 1 | 3 | 4 | 3
  Cycle 5 Day 1 Predose |  | 17.50 (NA) — GCV could not be calculated due to an insufficient number of participants available for analysis. | 30.79 (32) | 21.91 (109) | 33.64 (28)
  Cycle 5 Day 1 Postdose: number analyzed (Participants) | 0 | 1 | 2 | 4 | 3
  Cycle 5 Day 1 Postdose |  | 63.40 (NA) — GCV could not be calculated due to an insufficient number of participants available for analysis. | 102.03 (5) | 76.71 (29) | 98.97 (21)
  Cycle 6 Day 1 Predose: number analyzed (Participants) | 0 | 1 | 3 | 4 | 2
  Cycle 6 Day 1 Predose |  | 27.60 (NA) — GCV could not be calculated due to an insufficient number of participants available for analysis. | 24.08 (38) | 29.22 (74) | 40.73 (18)
  Cycle 9 Day 1 Predose: number analyzed (Participants) | 0 | 1 | 3 | 2 | 2
  Cycle 9 Day 1 Predose |  | 29.10 (NA) — GCV could not be calculated due to an insufficient number of participants available for analysis. | 36.28 (34) | 30.73 (34) | 37.67 (6)
  Cycle 13 Day 1 Predose: number analyzed (Participants) | 0 | 1 | 1 | 1 | 2
  Cycle 13 Day 1 Predose |  | 27.60 (NA) — GCV could not be calculated due to an insufficient number of participants available for analysis. | 36.70 (NA) — GCV could not be calculated due to an insufficient number of participants available for analysis. | 33.60 (NA) — GCV could not be calculated due to an insufficient number of participants available for analysis. | 25.02 (39)
  Cycle 17 Day 1 Predose: number analyzed (Participants) | 0 | 0 | 1 | 0 | 2
  Cycle 17 Day 1 Predose |  |  | 43.00 (NA) — GCV could not be calculated due to an insufficient number of participants available for analysis. |  | 26.79 (4)
  Cycle 25 Day 1 Predose: number analyzed (Participants) | 0 | 1 | 1 | 0 | 0
  Cycle 25 Day 1 Predose |  | 31.60 (NA) — GCV could not be calculated due to an insufficient number of participants available for analysis. | 56.20 (NA) — GCV could not be calculated due to an insufficient number of participants available for analysis. |  |

11. Secondary Outcome: Phase 1 (Dose Verification): Serum Concentrations of Ociperlimab
Description: Serum concentration of ociperlimab was determined. Post-dose refers to the data collected for 30 minutes post-infusion. "C" in the timeframe below refers to "Cycle" and D refers to "Day" and "h" refers to "hours".
Time Frame: Pre-dose, post-dose, 24 h,72 h,168 h,336 h post-dose C1D1, Pre-dose, post-dose on C2D1, Pre-dose, post-dose,168 h, 336 h post-dose on C5D1, Pre-dose, post-dose on C6D1, pre-dose C9D1 and C13D1 (each cycle = 21 days)
Population: Analysis was performed on PK Analysis set. Here, number analyzed' = participants with available data for the analysis of serum concentrations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Phase 1: Dose Verification: Cohort 1A (Ociperlimab 900 mg) | Phase 1: Dose Verification: Cohort 1B (Ociperlimab 900 mg + Tislelizumab 200 mg)
Number analyzed (Participants) | 9 | 11
micrograms per milliliter (mcg/mL)
  Cycle 1 Day 1- Predose | NA (NA) — Geometric mean and GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis. | NA (NA) — Geometric mean and GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis.
  Cycle 1 Day 1- Post-dose | 313.57 (21) | 267.78 (27)
  Cycle 1 Day 1- 24 h | 230.81 (29) | 201.98 (20)
  Cycle 1 Day 1- 72 h: number analyzed (Participants) | 8 | 11
  Cycle 1 Day 1- 72 h | 138.16 (43) | 141.37 (15)
  Cycle 1 Day 1- 168 h: number analyzed (Participants) | 8 | 11
  Cycle 1 Day 1- 168 h | 102.68 (27) | 99.84 (20)
  Cycle 1 Day 1- 336 h: number analyzed (Participants) | 8 | 9
  Cycle 1 Day 1- 336 h | 67.27 (52) | 59.10 (28)
  Cycle 2 Day 1- Pre-dose: number analyzed (Participants) | 7 | 9
  Cycle 2 Day 1- Pre-dose | 42.52 (58) | 30.53 (58)
  Cycle 2 Day 1- Post-dose: number analyzed (Participants) | 7 | 9
  Cycle 2 Day 1- Post-dose | 336.36 (24) | 316.63 (13)
  Cycle 5 Day 1- Pre-dose: number analyzed (Participants) | 1 | 3
  Cycle 5 Day 1- Pre-dose | 105.00 (NA) — GCV could not be calculated due to an insufficient number of participants available for analysis. | 43.02 (20)
  Cycle 5 Day 1- Post-dose: number analyzed (Participants) | 1 | 3
  Cycle 5 Day 1- Post-dose | 458.00 (NA) — GCV could not be calculated due to an insufficient number of participants available for analysis. | 360.55 (18)
  Cycle 5 Day 1- 168 h: number analyzed (Participants) | 1 | 3
  Cycle 5 Day 1- 168 h | 217.00 (NA) — GCV could not be calculated due to an insufficient number of participants available for analysis. | 126.19 (6)
  Cycle 5 Day 1- 336 h: number analyzed (Participants) | 1 | 3
  Cycle 5 Day 1- 336 h | 200.00 (NA) — GCV could not be calculated due to an insufficient number of participants available for analysis. | 76.09 (13)
  Cycle 6 Day 1- Pre-dose: number analyzed (Participants) | 1 | 3
  Cycle 6 Day 1- Pre-dose | 132.00 (NA) — GCV could not be calculated due to an insufficient number of participants available for analysis. | 53.96 (11)
  Cycle 6 Day 1- Post-dose: number analyzed (Participants) | 1 | 3
  Cycle 6 Day 1- Post-dose | 552.00 (NA) — GCV could not be calculated due to an insufficient number of participants available for analysis. | 355.69 (13)
  Cycle 9 Day 1- Pre-dose: number analyzed (Participants) | 1 | 2
  Cycle 9 Day 1- Pre-dose | 131.00 (NA) — GCV could not be calculated due to an insufficient number of participants available for analysis. | 66.92 (14)
  Cycle 13 Day 1- Pre-dose: number analyzed (Participants) | 1 | 1
  Cycle 13 Day 1- Pre-dose | 96.50 (NA) — GCV could not be calculated due to an insufficient number of participants available for analysis. | 61.30 (NA) — GCV could not be calculated due to an insufficient number of participants available for analysis.

12. Secondary Outcome: Phase 1 (Dose Verification): Serum Concentrations of Tislelizumab
Description: Serum concentrations of tislelizumab were determined. Post-dose refers to the data collected for 30 minutes post-infusion.
Time Frame: Cycle 1 Day 1 (pre-dose), Cycle 1 Day 1 (post-dose), Cycle 2 Day 1 (pre-dose), Cycle 5 Day 1 (pre-dose), Cycle 5 Day 1 (post-dose), Cycle 6 Day 1 (pre-dose), Cycle 9 Day 1 (pre-dose), Cycle 13 Day 1 (pre-dose) (each cycle = 21 days)
Population: Analysis was performed on PK Analysis set. Here number analyzed = participants with available data for analysis of serum concentrations. Data was not collected and analyzed for the "Phase 1: Dose Verification: Cohort 1A arm" because tislelizumab was not administered in that arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Phase 1: Dose Verification: Cohort 1B (Ociperlimab 900 mg + Tislelizumab 200 mg)
Number analyzed (Participants) | 11
micrograms per milliliter (mcg/mL)
  Cycle 1 Day 1- Pre-dose | NA (NA) — Geometric mean and GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis.
  Cycle 1 Day 1 Post-dose | 62.35 (26)
  Cycle 2 Day 1- Pre-dose: number analyzed (Participants) | 9
  Cycle 2 Day 1- Pre-dose | 14.67 (34)
  Cycle 5 Day 1- Pre-dose: number analyzed (Participants) | 3
  Cycle 5 Day 1- Pre-dose | 33.34 (22)
  Cycle 5 Day 1- Post-dose: number analyzed (Participants) | 3
  Cycle 5 Day 1- Post-dose | 117.68 (9)
  Cycle 6 Day 1- Pre-dose: number analyzed (Participants) | 3
  Cycle 6 Day 1- Pre-dose | 36.41 (4)
  Cycle 9 Day 1- Pre-dose: number analyzed (Participants) | 2
  Cycle 9 Day 1- Pre-dose | 46.76 (6)
  Cycle 13 Day 1- Pre-dose: number analyzed (Participants) | 1
  Cycle 13 Day 1- Pre-dose | 48.30 (NA) — GCV could not be calculated due to an insufficient number of participants available for analysis.

13. Secondary Outcome: Phase 1: Number of Participants With Immunogenic Response to Ociperlimab and Tislelizumab
Description: Immunogenic responses to ociperlimab and tislelizumab included: treatment emergent, treatment-induced and treatment boosted anti-drug antibodies (ADA) and neutralizing antibody (NAb) positive assessments. Treatment-emergent ADA was defined as the sum of treatment-boosted ADA and treatment-induced ADA participants. Treatment-induced ADA was defined as ADA-evaluable participants that were ADA-negative at baseline and ADA-positive after drug administration during the treatment or follow-up observation period. Treatment-boosted ADA was defined as the Baseline-positive ADA-evaluable participants with significant increases (4-fold or higher) in ADA titer after drug administration during the treatment or follow-up observation period. NAb positive was defined as ADA-evaluable participants with positive Nab at any time including baseline and/or after drug administration.
Time Frame: Up to 32.2 months (Dose escalation cohorts) and up to 11 months (Dose verification cohorts)
Population: Analysis was performed on ADA Analysis Set that included all participants who received at least 1 dose of any component of study drugs for whom both baseline antidrug antibody result and at least 1 corresponding post-baseline antidrug antibody result are available. Here, number analyzed = participants with available data for the ADA analysis and "0" in the number analyzed signifies no participant were available for analysis at specified time-points.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Dose Escalation: Ociperlimab 50 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 150 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 450 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 900 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 1800 mg + Tislelizumab 200 mg | Phase 1: Dose Verification: Cohort 1A (Ociperlimab 900 mg) | Phase 1: Dose Verification: Cohort 1B (Ociperlimab 900 mg + Tislelizumab 200 mg)
Number analyzed (Participants) | 1 | 3 | 6 | 16 | 6 | 9 | 11
Participants
  Ociperlimab: Treatment-Emergent ADAs: number analyzed (Participants) | 1 | 3 | 6 | 14 | 5 | 8 | 9
  Ociperlimab: Treatment-Emergent ADAs | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ociperlimab: Treatment-Induced ADAs: number analyzed (Participants) | 1 | 3 | 6 | 14 | 5 | 8 | 9
  Ociperlimab: Treatment-Induced ADAs | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ociperlimab: Treatment-Boosted ADAs: number analyzed (Participants) | 1 | 3 | 6 | 14 | 5 | 8 | 9
  Ociperlimab: Treatment-Boosted ADAs | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ociperlimab: NAb Positive: number analyzed (Participants) | 1 | 3 | 6 | 14 | 5 | 8 | 9
  Ociperlimab: NAb Positive | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Tislelizumab: Treatment-Emergent ADAs: number analyzed (Participants) | 1 | 3 | 6 | 14 | 5 | 0 | 9
  Tislelizumab: Treatment-Emergent ADAs | 1 | 0 | 2 | 1 | 1 |  | 2
  Tislelizumab: Treatment-Induced ADAs: number analyzed (Participants) | 1 | 3 | 6 | 14 | 5 | 0 | 9
  Tislelizumab: Treatment-Induced ADAs | 1 | 0 | 2 | 1 | 1 |  | 1
  Tislelizumab: Treatment-Boosted ADAs: number analyzed (Participants) | 1 | 3 | 6 | 14 | 5 | 0 | 9
  Tislelizumab: Treatment-Boosted ADAs | 0 | 0 | 0 | 0 | 0 |  | 1
  Tislelizumab: NAb Positive: number analyzed (Participants) | 1 | 3 | 6 | 14 | 5 | 0 | 9
  Tislelizumab: NAb Positive | 0 | 0 | 0 | 0 | 0 |  | 0

14. Secondary Outcome: Phase 1b: DOR as Per RECIST v.1.1
Description: DOR was defined as the time from the first determination of an overall response per RECIST v1.1 until the first documentation of progression or death, whichever came first. DOR was estimated using the Kaplan-Meier method. Per RECIST v.1.1., CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study.
Time Frame: From the first determination of an overall response until PD or death, whichever came first (Maximum time duration on study: Up to 41.6 months [Cohorts 1 to 9] and up to 21.4 months [Cohort 10])
Population: Analysis was performed on participants in efficacy evaluable analysis set with an objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b: Dose Expansion: Cohort 1 | Phase 1b: Dose Expansion: Cohort 2 | Phase 1b: Dose Expansion: Cohort 3 | Phase 1b: Dose Expansion: Cohort 4 | Phase 1b: Dose Expansion: Cohort 5 | Phase 1b: Dose Expansion: Cohort 6 | Phase 1b: Dose Expansion: Cohort 7 | Phase 1b: Dose Expansion: Cohort 8 | Phase 1b: Dose Expansion: Cohort 9 | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 450 mg + Tislelizumab 200 mg) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 900 mg + Tislelizumab 200 mg) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 1800 mg + Tislelizumab 200 mg)
Number analyzed (Participants) | 22 | 23 | 18 | 27 | 2 | 13 | 2 | 13 | 30 | 8 | 5 | 8
months | 16.9 [5.6 to NA] — Upper limit of 95% CI could not be calculated due to an insufficient number of participants with a response. | 13.9 [8.2 to NA] — Upper limit of 95% CI could not be calculated due to an insufficient number of participants with a response. | 14.0 [2.9 to NA] — Upper limit of 95% CI could not be calculated due to an insufficient number of participants with a response. | 4.1 [3.4 to 5.6] | 15.9 [12.6 to NA] — Upper limit of 95% CI could not be calculated due to an insufficient number of participants with a response. | 8.0 [5.3 to 10.9] | 3.4 [2.1 to NA] — Upper limit of 95% CI could not be calculated due to an insufficient number of participants with a response. | 8.5 [2.8 to NA] — Upper limit of 95% CI could not be calculated due to an insufficient number of participants with a response. | 8.4 [5.6 to 13.4] | 16.6 [3.9 to NA] — Upper limit of 95% CI could not be calculated due to an insufficient number of participants with a response. | NA [6.3 to NA] — Median and upper limit of 95% CI could not be calculated due to an insufficient number of participants with a response. | 8.3 [5.3 to NA] — Upper limit of 95% CI could not be calculated due to an insufficient number of participants with a response.

15. Secondary Outcome: Phase 1b: DCR as Per RECIST v.1.1
Description: DCR was defined as the percentage of participants with BOR, as per RECIST v.1.1, of a CR, PR, or SD. Per Response evaluation criteria in solid tumors (RECIST) version (v)1.1., CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: as for outcome 14
Population: Analysis was performed on efficacy evaluable analysis set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase 1b: Dose Expansion: Cohort 9: Participants with unresectable, locally advanced, recurrent, or metastatic G/GEJ adenocarcinoma received treatment with 6 cycles of ociperlimab 900 mg (Day 1) IV infusion, tislelizumab 200 mg (Day 1) IV infusion, (oxaliplatin 1300 mg/m^2 [Day 1] and capecitabine 1000 mg/m^2 [Day 1-14 twice daily], or cisplatin 75 mg/m^2 [Day], and 5-FU 750-800 mg/m^2 [Day 1-5]) Q3W followed by ociperlimab 900 mg (Day 1), tislelizumab 200 mg (Day 1) + capecitabine 1000 mg/m^2 twice daily (Day 1-14) Q3W until disease progression, intolerable toxicity, or withdrawal of consent.
Arm/Group | Phase 1b: Dose Expansion: Cohort 1 | Phase 1b: Dose Expansion: Cohort 2 | Phase 1b: Dose Expansion: Cohort 3 | Phase 1b: Dose Expansion: Cohort 4 | Phase 1b: Dose Expansion: Cohort 5 | Phase 1b: Dose Expansion: Cohort 6 | Phase 1b: Dose Expansion: Cohort 7 | Phase 1b: Dose Expansion: Cohort 8 | Phase 1b: Dose Expansion: Cohort 9 | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 450 mg + Tislelizumab 200 mg) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 900 mg + Tislelizumab 200 mg) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 1800 mg + Tislelizumab 200 mg)
Number analyzed (Participants) | 40 | 42 | 45 | 41 | 26 | 19 | 6 | 39 | 59 | 23 | 19 | 23
percentage of participants | 90.0 [76.3 to 97.2] | 92.9 [80.5 to 98.5] | 86.7 [73.2 to 94.9] | 90.2 [76.9 to 97.3] | 53.8 [33.4 to 73.4] | 94.7 [74.0 to 99.9] | 83.3 [35.9 to 99.6] | 69.2 [52.4 to 83.0] | 86.4 [75.0 to 94.0] | 34.8 [16.4 to 57.3] | 26.3 [9.1 to 51.2] | 34.8 [16.4 to 57.3]

16. Secondary Outcome: Phase 1b: Progression Free Survival (PFS) as Per RECIST v.1.1
Description: PFS was defined as the time from the date of the first dose of study drugs to the date of the first documentation of PD assessed by the investigator using RECIST v1.1 or death, whichever occurred first. PFS was estimated using the Kaplan-Meier method. Per RECIST v1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study.
Time Frame: From first dose of study drugs to the date of the first documentation of PD or death, whichever came first (Maximum time duration on study: up to 41.6 months [Cohorts 1 to 9] and up to 21.4 months [Cohort 10])
Population: Analysis was performed on safety analysis set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b: Dose Expansion: Cohort 1 | Phase 1b: Dose Expansion: Cohort 2 | Phase 1b: Dose Expansion: Cohort 3 | Phase 1b: Dose Expansion: Cohort 4 | Phase 1b: Dose Expansion: Cohort 5 | Phase 1b: Dose Expansion: Cohort 6 | Phase 1b: Dose Expansion: Cohort 7 | Phase 1b: Dose Expansion: Cohort 8 | Phase 1b: Dose Expansion: Cohort 9 | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 450 mg + Tislelizumab 200 mg) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 900 mg + Tislelizumab 200 mg) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 1800 mg + Tislelizumab 200 mg)
Number analyzed (Participants) | 41 | 43 | 45 | 43 | 26 | 21 | 6 | 41 | 60 | 24 | 21 | 23
months | 8.2 [6.0 to 18.1] | 11.3 [8.0 to 20.7] | 5.5 [4.2 to 8.2] | 4.9 [4.2 to 5.5] | 2.9 [1.4 to 5.3] | 7.9 [4.1 to 10.7] | 4.9 [2.0 to NA] — Upper limit of 95% CI could not be calculated due to an insufficient number of participants with events. | 5.7 [3.0 to 8.3] | 7.3 [5.1 to 9.5] | 2.8 [1.4 to 6.8] | 1.9 [1.2 to 9.0] | 8.2 [5.5 to 11.0]

17. Secondary Outcome: Phase 1b (Cohorts 1-10): Number of Participants With TEAEs and TESAEs
Description: An AE was defined as any unfavorable and unintended sign, symptom, or disease associated with the use of study drugs, whether considered related to study drugs or not. An SAE was any untoward medical occurrence that, at any dose, resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability, was a congenital anomaly or was considered a medically significant. TEAE was an AE that has an onset date or a worsening in severity from baseline on or after the first dose of study drug up to 30 days following study drug discontinuation or initiation of the first new systemic anticancer therapy, whichever occurred first. Severity of AEs was assessed according to NCI-CTCAE v.5.0, which consists of: Grade 1 Mild; Grade 2 Moderate; Grade 3: Severe; Grade 4: Life-threatening; Grade 5: Death due to AE.
Time Frame: Up to 30 days after the last dose of study interventions (Maximum time duration on study: up to 41.6 months [Cohorts 1 to 9] and up to 21.4 months [Cohort 10])
Population: Analysis was performed on safety set.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Dose Expansion: Cohort 1 | Phase 1b: Dose Expansion: Cohort 2 | Phase 1b: Dose Expansion: Cohort 3 | Phase 1b: Dose Expansion: Cohort 4 | Phase 1b: Dose Expansion: Cohort 5 | Phase 1b: Dose Expansion: Cohort 6 | Phase 1b: Dose Expansion: Cohort 7 | Phase 1b: Dose Expansion: Cohort 8 | Phase 1b: Dose Expansion: Cohort 9 | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 450 mg + Tislelizumab 200 mg) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 900 mg + Tislelizumab 200 mg) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 1800 mg + Tislelizumab 200 mg)
Number analyzed (Participants) | 41 | 43 | 45 | 43 | 26 | 21 | 6 | 41 | 60 | 24 | 21 | 23
Participants
  Participants with any TEAE | 41 | 43 | 44 | 43 | 25 | 21 | 6 | 41 | 60 | 23 | 18 | 23
  Participants with >= Grade 3 TEAE | 30 | 33 | 17 | 31 | 12 | 16 | 6 | 27 | 49 | 9 | 10 | 15
  Serious TEAE | 21 | 28 | 15 | 23 | 9 | 11 | 4 | 22 | 32 | 10 | 8 | 13

18. Secondary Outcome: Phase 1b (Cohort 1-9): Serum Concentrations of Ociperlimab
Description: Serum concentrations of ociperlimab were determined. Post-dose refers to the data collected for 30 minutes post-infusion.
Time Frame: Cycle 1 Day 1 (pre-dose), Cycle 1 Day 1 (post-dose), Cycle 2 Day 1 (pre-dose), Cycle 5 Day 1 (pre-dose and post-dose), pre-dose on Cycle 6 Day 1, Cycle 9 Day 1, Cycle 13 Day 1, Cycle 17 Day 1 and Cycle 25 Day 1 (each cycle = 21 days)
Population: Analysis was performed on PK analysis set. Here, "Overall number of participants analyzed" = participants with available data for this outcome measure and 'number analyzed' = the number of participants with available data for the analysis of serum concentrations and "0" in the number analyzed signifies no participant with available data at specified time-points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (mcg/mL)
Groups:
- Phase 1b: Dose Expansion: Cohort 2: Participants with metastatic non-squamous NSCLC (PD-L1 positive, TC >= 1%) received treatment with ociperlimab 900 mg IV infusion and tislelizumab 200 mg IV infusion on Day 1 of each 21-day cycle. Participants also received cisplatin 75 mg/m^2 or carboplatin (AUC 5) and pemetrexed 500 mg/m^2 (on Day 1) Q3W for 4-6 cycles followed by ociperlimab 900 mg + tislelizumab 200 mg + pemetrexed 500 mg/m^2 on Day 1 Q3W until disease progression, intolerable toxicity, or withdrawal of consent.
Arm/Group | Phase 1b: Dose Expansion: Cohort 1 | Phase 1b: Dose Expansion: Cohort 2 | Phase 1b: Dose Expansion: Cohort 3 | Phase 1b: Dose Expansion: Cohort 4 | Phase 1b: Dose Expansion: Cohort 5 | Phase 1b: Dose Expansion: Cohort 6 | Phase 1b: Dose Expansion: Cohort 7 | Phase 1b: Dose Expansion: Cohort 8 | Phase 1b: Dose Expansion: Cohort 9
Number analyzed (Participants) | 41 | 43 | 45 | 43 | 26 | 21 | 6 | 41 | 59
micrograms per milliliter (mcg/mL)
  Cycle 1 Day 1-Pre-dose: number analyzed (Participants) | 41 | 42 | 45 | 43 | 26 | 21 | 5 | 41 | 58
  Cycle 1 Day 1-Pre-dose | NA (NA) — Geometric mean and GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis. | NA (NA) — Geometric mean and GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis. | NA (NA) — Geometric mean and GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis. | NA (NA) — Geometric mean and GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis. | NA (NA) — Geometric mean and GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis. | NA (NA) — Geometric mean and GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis. | NA (NA) — Geometric mean and GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis. | NA (NA) — Geometric mean and GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis. | NA (NA) — Geometric mean and GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis.
  Cycle 1 Day 1- Post-dose: number analyzed (Participants) | 41 | 41 | 44 | 41 | 21 | 20 | 4 | 41 | 57
  Cycle 1 Day 1- Post-dose | 293.20 (30) | 296.90 (24) | 287.70 (23) | 282.22 (28) | 259.50 (30) | 295.38 (30) | 212.61 (23) | 308.25 (27) | 251.33 (27)
  Cycle 2 Day 1- Pre-dose: number analyzed (Participants) | 35 | 38 | 41 | 38 | 23 | 18 | 5 | 35 | 52
  Cycle 2 Day 1- Pre-dose | 32.06 (51) | 35.93 (62) | 32.63 (55) | 34.69 (38) | 30.98 (101) | 33.09 (52) | 19.74 (249) | 37.52 (62) | 32.52 (53)
  Cycle 5 Day 1- Pre-dose: number analyzed (Participants) | 32 | 31 | 27 | 32 | 9 | 15 | 4 | 23 | 37
  Cycle 5 Day 1- Pre-dose | 70.55 (50) | 80.94 (75) | 65.66 (64) | 72.81 (42) | 79.91 (86) | 90.20 (34) | 69.98 (62) | 67.90 (100) | 70.39 (46)
  Cycle 5 Day 1- Post-dose: number analyzed (Participants) | 32 | 30 | 26 | 30 | 10 | 15 | 4 | 23 | 36
  Cycle 5 Day 1- Post-dose | 386.03 (25) | 382.09 (23) | 354.15 (21) | 344.61 (24) | 329.26 (20) | 338.17 (22) | 327.12 (29) | 391.94 (25) | 324.40 (31)
  Cycle 6 Day 1- Pre-dose: number analyzed (Participants) | 32 | 27 | 28 | 28 | 8 | 15 | 2 | 20 | 35
  Cycle 6 Day 1- Pre-dose | 77.56 (51) | 88.71 (60) | 68.12 (59) | 77.98 (47) | 88.08 (85) | 74.72 (102) | 127.53 (25) | 77.27 (78) | 68.02 (73)
  Cycle 9 Day 1- Pre-dose: number analyzed (Participants) | 22 | 27 | 17 | 15 | 6 | 9 | 2 | 16 | 27
  Cycle 9 Day 1- Pre-dose | 78.12 (68) | 103.40 (61) | 78.16 (44) | 85.51 (49) | 101.98 (87) | 85.98 (48) | 171.57 (38) | 94.91 (68) | 73.16 (88)
  Cycle 13 Day 1- Pre-dose: number analyzed (Participants) | 17 | 21 | 9 | 9 | 4 | 9 | 0 | 12 | 19
  Cycle 13 Day 1- Pre-dose | 98.90 (35) | 112.33 (66) | 90.14 (48) | 92.58 (34) | 76.79 (65) | 85.49 (61) |  | 105.69 (74) | 94.79 (58)
  Cycle 17 Day 1- Pre-dose: number analyzed (Participants) | 13 | 13 | 8 | 4 | 3 | 3 | 0 | 7 | 9
  Cycle 17 Day 1- Pre-dose | 89.49 (45) | 111.36 (43) | 91.84 (39) | 93.32 (68) | 14.78 (6698) | 78.30 (9) |  | 104.02 (76) | 101.27 (66)
  Cycle 25 Day 1- Pre-dose: number analyzed (Participants) | 12 | 13 | 7 | 4 | 2 | 1 | 0 | 0 | 3
  Cycle 25 Day 1- Pre-dose | 102.28 (35) | 120.07 (37) | 85.34 (47) | 97.04 (51) | 72.98 (85) | 56.00 (NA) — GCV could not be calculated due to an insufficient number of participants available for analysis. |  |  | 58.44 (96)

19. Secondary Outcome: Phase 1b (Cohort 1-9): Serum Concentrations of Tislelizumab
Description: as for outcome 12
Time Frame: Cycle 1 Day 1 (pre-dose and post-dose), Cycle 2 Day 1 (pre-dose), Cycle 5 Day 1 (pre-dose and post-dose), pre-dose on Cycle 6 Day 1, Cycle 9 Day 1, Cycle 13 Day 1, Cycle 17 Day 1 and Cycle 25 Day 1 (each cycle = 21 days)
Population: Analysis was performed on PK analysis set. Here, number analyzed' = participants with available data for the analysis of serum concentrations and "0" in the number analyzed signifies no participant with available data at specified time-points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Phase 1b: Dose Expansion: Cohort 1 | Phase 1b: Dose Expansion: Cohort 2 | Phase 1b: Dose Expansion: Cohort 3 | Phase 1b: Dose Expansion: Cohort 4 | Phase 1b: Dose Expansion: Cohort 5 | Phase 1b: Dose Expansion: Cohort 6 | Phase 1b: Dose Expansion: Cohort 7 | Phase 1b: Dose Expansion: Cohort 8 | Phase 1b: Dose Expansion: Cohort 9
Number analyzed (Participants) | 41 | 43 | 45 | 43 | 26 | 21 | 6 | 41 | 60
micrograms per milliliter (mcg/mL)
  Cycle 1 Day 1-Pre-dose: number analyzed (Participants) | 41 | 42 | 45 | 43 | 25 | 21 | 6 | 41 | 59
  Cycle 1 Day 1-Pre-dose | 2.13 (NA) — GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis. | 45.40 (NA) — GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis. | 35.20 (NA) — GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis. | 1.35 (NA) — GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis. | 25.78 (NA) — GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis. | 36.00 (NA) — GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis. | NA (NA) — Geometric mean and GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis. | NA (NA) — Geometric mean and GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis. | NA (NA) — Geometric mean and GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis.
  Cycle 1 Day 1-Post-dose: number analyzed (Participants) | 41 | 42 | 44 | 42 | 22 | 19 | 5 | 41 | 58
  Cycle 1 Day 1-Post-dose | 68.69 (19) | 70.24 (21) | 70.07 (21) | 65.59 (27) | 86.72 (28) | 65.15 (22) | 52.88 (11) | 69.50 (19) | 59.14 (23)
  Cycle 2 Day 1-Pre-dose: number analyzed (Participants) | 35 | 38 | 41 | 38 | 23 | 18 | 5 | 35 | 52
  Cycle 2 Day 1-Pre-dose | 16.16 (33) | 17.22 (48) | 16.51 (32) | 17.00 (32) | 29.46 (59) | 14.31 (35) | 12.58 (36) | 17.33 (41) | 13.91 (38)
  Cycle 5 Day 1-Pre-dose: number analyzed (Participants) | 33 | 30 | 27 | 33 | 9 | 15 | 4 | 23 | 37
  Cycle 5 Day 1-Pre-dose | 36.32 (43) | 35.45 (98) | 31.50 (65) | 38.54 (35) | 36.32 (46) | 39.78 (22) | 28.96 (50) | 37.33 (67) | 29.46 (48)
  Cycle 5 Day 1-Post-dose: number analyzed (Participants) | 33 | 29 | 26 | 31 | 10 | 15 | 4 | 23 | 35
  Cycle 5 Day 1-Post-dose | 105.78 (28) | 107.03 (29) | 105.03 (24) | 104.12 (23) | 100.39 (20) | 97.03 (24) | 72.73 (26) | 109.71 (28) | 86.46 (27)
  Cycle 6 Day 1-Pre-dose: number analyzed (Participants) | 32 | 27 | 28 | 28 | 8 | 14 | 2 | 20 | 35
  Cycle 6 Day 1-Pre-dose | 38.56 (40) | 37.47 (95) | 34.48 (47) | 39.78 (36) | 39.30 (47) | 36.91 (93) | 44.63 (47) | 43.60 (48) | 29.37 (64)
  Cycle 9 Day 1-Pre-dose: number analyzed (Participants) | 22 | 27 | 17 | 15 | 6 | 9 | 2 | 16 | 27
  Cycle 9 Day 1-Pre-dose | 40.32 (54) | 37.29 (128) | 40.98 (45) | 47.24 (29) | 42.50 (53) | 40.62 (48) | 63.54 (77) | 48.29 (51) | 27.03 (138)
  Cycle 13 Day 1-Pre-dose: number analyzed (Participants) | 17 | 21 | 9 | 9 | 4 | 9 | 0 | 12 | 19
  Cycle 13 Day 1-Pre-dose | 48.48 (35) | 47.22 (42) | 43.46 (28) | 51.62 (16) | 45.87 (59) | 38.19 (30) |  | 47.08 (70) | 36.61 (75)
  Cycle 17 Day 1-Pre-dose: number analyzed (Participants) | 13 | 13 | 8 | 4 | 3 | 3 | 0 | 7 | 9
  Cycle 17 Day 1-Pre-dose | 46.36 (35) | 48.39 (29) | 46.91 (20) | 48.96 (55) | 51.48 (11) | 36.71 (10) |  | 48.23 (68) | 40.14 (86)
  Cycle 25 Day 1-Pre-dose: number analyzed (Participants) | 12 | 13 | 7 | 4 | 2 | 1 | 0 | 0 | 3
  Cycle 25 Day 1-Pre-dose | 48.48 (25) | 52.34 (26) | 44.47 (30) | 49.65 (40) | 42.97 (35) | 21.40 (NA) — GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis. |  |  | 16.83 (117)

20. Secondary Outcome: Phase 1b (Cohort 10): Serum Concentrations of Ociperlimab
Description: Serum concentrations of ociperlimab were determined. Post-dose refers to the data collected for 30 minutes post-infusion and 'h' in the time-frame section refers to hours.
Time Frame: Pre-dose, post-dose, 168 h, 336 h post-dose Cycle1 Day 1, Pre-dose on Cycle 2 Day 1, Pre-dose, post-dose (30 min) on Cycle 5 Day 1, Pre-dose on Cycle 6 Day 1, Cycle 9 Day 1, Cycle 13 Day 1, Cycle 17 Day 1, and Cycle 25 Day 1 (each cycle = 21 days)
Population: Analysis was performed on PK analysis set. Here, 'number analyzed' = participants with available data for the analysis of serum concentrations and "0" in the number analyzed signifies that no participant with available data at the specified time-point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 450 mg + Tislelizumab 200 mg) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 900 mg + Tislelizumab 200 mg) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 1800 mg + Tislelizumab 200 mg)
Number analyzed (Participants) | 24 | 21 | 23
micrograms per milliliter (mcg/mL)
  Cycle 1 Day 1- Pre-dose | NA (NA) — Geometric mean and GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis. | NA (NA) — Geometric mean and GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis. | NA (NA) — Geometric mean and GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis.
  Cycle 1 Day 1- Post-dose: number analyzed (Participants) | 24 | 20 | 21
  Cycle 1 Day 1- Post-dose | 147.73 (21) | 309.74 (15) | 580.37 (15)
  Cycle 1 Day 1- 168 h: number analyzed (Participants) | 22 | 18 | 19
  Cycle 1 Day 1- 168 h | 44.61 (32) | 99.03 (25) | 178.34 (26)
  Cycle 1 Day 1- 336 h: number analyzed (Participants) | 22 | 18 | 20
  Cycle 1 Day 1- 336 h | 25.65 (41) | 56.73 (49) | 103.48 (31)
  Cycle 2 Day 1- Pre-dose: number analyzed (Participants) | 20 | 17 | 19
  Cycle 2 Day 1- Pre-dose | 13.02 (66) | 31.60 (49) | 64.10 (33)
  Cycle 5 Day 1- Pre-dose: number analyzed (Participants) | 9 | 10 | 18
  Cycle 5 Day 1- Pre-dose | 40.02 (54) | 67.49 (49) | 95.90 (82)
  Cycle 5 Day 1- Post-dose: number analyzed (Participants) | 9 | 10 | 18
  Cycle 5 Day 1- Post-dose | 217.47 (16) | 404.63 (20) | 664.37 (13)
  Cycle 6 Day 1- Pre-dose: number analyzed (Participants) | 9 | 10 | 16
  Cycle 6 Day 1- Pre-dose | 27.74 (331) | 68.08 (54) | 110.97 (45)
  Cycle 9 Day 1- Pre-dose: number analyzed (Participants) | 5 | 7 | 13
  Cycle 9 Day 1- Pre-dose | 55.13 (31) | 86.59 (95) | 89.60 (166)
  Cycle 13 Day 1- Pre-dose: number analyzed (Participants) | 2 | 6 | 6
  Cycle 13 Day 1- Pre-dose | 61.11 (41) | 86.89 (32) | 142.18 (36)
  Cycle 17 Day 1- Pre-dose: number analyzed (Participants) | 3 | 3 | 3
  Cycle 17 Day 1- Pre-dose | 52.56 (22) | 105.58 (23) | 119.15 (21)
  Cycle 25 Day 1- Pre-dose: number analyzed (Participants) | 1 | 0 | 1
  Cycle 25 Day 1- Pre-dose | 108.00 (NA) — GCV could not be calculated due to an insufficient number of participants available for analysis. |  | 125.00 (NA) — GCV could not be calculated due to an insufficient number of participants available for analysis.

21. Secondary Outcome: Phase 1b (Cohort 10): Serum Concentrations of Tislelizumab
Description: as for outcome 12
Time Frame: Cycle 1 Day 1 (pre-dose and post-dose, Cycle 2 Day 1 (pre-dose), Cycle 5 Day 1 (pre-dose and post-dose), pre-dose of Cycle 6 Day 1, Cycle 9 Day 1, Cycle 13 Day 1, Cycle 17 Day 1 and Cycle 25 Day 1 (each cycle = 21 days)
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 450 mg + Tislelizumab 200 mg) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 900 mg + Tislelizumab 200 mg) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 1800 mg + Tislelizumab 200 mg)
Number analyzed (Participants) | 24 | 21 | 23
micrograms per milliliter (mcg/mL)
  Cycle 1 Day 1-Pre-dose | NA (NA) — Geometric mean and GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis. | 2.94 (317) | NA (NA) — Geometric mean and GCV could not be calculated due to an insufficient number of participants with LLOQ for analysis.
  Cycle 1 Day 1-Post-dose: number analyzed (Participants) | 24 | 20 | 22
  Cycle 1 Day 1-Post-dose | 68.42 (24) | 67.97 (12) | 63.62 (17)
  Cycle 2 Day 1-Pre-dose: number analyzed (Participants) | 20 | 17 | 19
  Cycle 2 Day 1-Pre-dose | 13.81 (45) | 14.87 (31) | 14.70 (32)
  Cycle 5 Day 1-Pre-dose: number analyzed (Participants) | 9 | 10 | 18
  Cycle 5 Day 1-Pre-dose | 36.10 (43) | 35.56 (34) | 25.24 (52)
  Cycle 5 Day 1-Post-dose: number analyzed (Participants) | 9 | 10 | 18
  Cycle 5 Day 1-Post-dose | 117.14 (27) | 103.69 (16) | 90.46 (17)
  Cycle 6 Day 1-Pre-dose: number analyzed (Participants) | 9 | 10 | 16
  Cycle 6 Day 1-Pre-dose | 34.73 (80) | 35.17 (34) | 28.70 (39)
  Cycle 9 Day 1-Pre-dose: number analyzed (Participants) | 5 | 7 | 13
  Cycle 9 Day 1-Pre-dose | 53.01 (29) | 48.07 (64) | 25.96 (110)
  Cycle 13 Day 1-Pre-dose: number analyzed (Participants) | 2 | 6 | 6
  Cycle 13 Day 1-Pre-dose | 73.38 (19) | 42.67 (36) | 37.52 (20)
  Cycle 17 Day 1-Pre-dose: number analyzed (Participants) | 3 | 3 | 3
  Cycle 17 Day 1-Pre-dose | 59.21 (13) | 55.86 (18) | 29.99 (40)
  Cycle 25 Day 1-Pre-dose: number analyzed (Participants) | 1 | 0 | 1
  Cycle 25 Day 1-Pre-dose | 82.30 (NA) — GCV could not be calculated due to an insufficient number of participants available for analysis. |  | 32.80 (NA) — GCV could not be calculated due to an insufficient number of participants available for analysis.

22. Secondary Outcome: Phase 1b (Cohort 1-10): Number of Participants With Immunogenic Response to Ociperlimab and Tislelizumab
Description: Immunogenic responses to ociperlimab and tislelizumab included: treatment emergent, treatment-induced and treatment boosted ADA and NAb positive assessments. Treatment-emergent ADA was defined as the sum of treatment-boosted ADA and treatment-induced ADA participants. Treatment-induced ADA was defined as ADA-evaluable participants that were ADA-negative at baseline and ADA-positive after drug administration during the treatment or follow-up observation period. Treatment-boosted ADA was defined as the Baseline-positive ADA-evaluable participants with significant increases (4-fold or higher) in ADA titer after drug administration during the treatment or follow-up observation period. NAb positive was defined as ADA-evaluable participants with positive Nab at any time including baseline and/or after drug administration.
Time Frame: Up to 34.4 months (Cohorts 1 to 9) and up to 20.8 months (Cohort 10)
Population: Analysis was performed on ADA Analysis set. Here, number analyzed = participants with available data for ADA analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Dose Expansion: Cohort 1 | Phase 1b: Dose Expansion: Cohort 2 | Phase 1b: Dose Expansion: Cohort 3 | Phase 1b: Dose Expansion: Cohort 4 | Phase 1b: Dose Expansion: Cohort 5 | Phase 1b: Dose Expansion: Cohort 6 | Phase 1b: Dose Expansion: Cohort 7 | Phase 1b: Dose Expansion: Cohort 8 | Phase 1b: Dose Expansion: Cohort 9 | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 450 mg + Tislelizumab 200 mg) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 900 mg + Tislelizumab 200 mg) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 1800 mg + Tislelizumab 200 mg)
Number analyzed (Participants) | 41 | 43 | 45 | 43 | 26 | 21 | 6 | 41 | 60 | 24 | 21 | 23
Participants
  Ociperlimab: Treatment-Emergent ADAs: number analyzed (Participants) | 37 | 41 | 44 | 40 | 25 | 18 | 5 | 37 | 53 | 21 | 18 | 21
  Ociperlimab: Treatment-Emergent ADAs | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ociperlimab: Treatment-Boosted ADAs: number analyzed (Participants) | 37 | 41 | 44 | 40 | 25 | 18 | 5 | 37 | 53 | 21 | 18 | 21
  Ociperlimab: Treatment-Boosted ADAs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ociperlimab: Treatment-Induced ADAs: number analyzed (Participants) | 37 | 41 | 44 | 40 | 25 | 18 | 5 | 37 | 53 | 21 | 18 | 21
  Ociperlimab: Treatment-Induced ADAs | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ociperlimab NAb positive: number analyzed (Participants) | 37 | 41 | 44 | 40 | 25 | 18 | 5 | 37 | 53 | 21 | 18 | 21
  Ociperlimab NAb positive | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Tislelizumab: Treatment-Emergent ADAs: number analyzed (Participants) | 37 | 41 | 44 | 40 | 24 | 18 | 5 | 37 | 53 | 21 | 18 | 21
  Tislelizumab: Treatment-Emergent ADAs | 24 | 17 | 17 | 12 | 3 | 11 | 2 | 10 | 17 | 11 | 6 | 9
  Tislelizumab: Treatment-Boosted ADAs: number analyzed (Participants) | 37 | 41 | 44 | 40 | 24 | 18 | 5 | 37 | 53 | 21 | 18 | 21
  Tislelizumab: Treatment-Boosted ADAs | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0
  Tislelizumab: Treatment-Induced ADAs: number analyzed (Participants) | 37 | 41 | 44 | 40 | 24 | 18 | 5 | 37 | 53 | 21 | 18 | 21
  Tislelizumab: Treatment-Induced ADAs | 22 | 16 | 16 | 11 | 3 | 11 | 2 | 9 | 17 | 9 | 5 | 9
  Tislelizumab NAb positive: number analyzed (Participants) | 37 | 41 | 44 | 40 | 24 | 18 | 5 | 37 | 53 | 21 | 18 | 21
  Tislelizumab NAb positive | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

23. Secondary Outcome: Phase 1b (Cohort 1-10): Percentage of Participants With ORR: TIGIT Biomarkers Expression
Description: Archival or fresh tumor samples were collected for analysis of biomarkers for T cell immunoglobulin and immunoreceptor tyrosine-based inhibitory motif (ITIM) domain (TIGIT) and PD-L1 expression.
  The TIGIT expression on immune cells (IC) and the classification thresholds were different for various cohorts. For Cohort 4, TIGIT IC was categorized as <1% or >=1%; for Cohorts 1, 2, 3, 5, 6, 8, 9 and 10, TIGIT IC was categorized as <5% or >=5%.
  ORR is reported for each TIGIT subgroup as relevant in each cohort. Biomarker data were not analyzed and reported for participants in Cohort 7.
Time Frame: Maximum time duration on study: up to 41.6 months (Cohorts 1 to 9) and up to 21.4 months (Cohort 10)
Population: Analysis was performed on efficacy evaluable analysis set for participants with available TIGIT or PD-L1 expression levels. Here, "Overall number of participants analyzed" = participants with available data for this outcome measure and "number analyzed" signifies participants with available data for each specified category at respective visit and "0" in the number analyzed defines no participant were available for analysis at specified time-points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1b: Dose Expansion: Cohort 1 | Phase 1b: Dose Expansion: Cohort 2 | Phase 1b: Dose Expansion: Cohort 3 | Phase 1b: Dose Expansion: Cohort 4 | Phase 1b: Dose Expansion: Cohort 5 | Phase 1b: Dose Expansion: Cohort 6 | Phase 1b: Dose Expansion: Cohort 7 | Phase 1b: Dose Expansion: Cohort 8 | Phase 1b: Dose Expansion: Cohort 9 | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 450 mg + Tislelizumab 200 mg) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 900 mg + Tislelizumab 200 mg) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 1800 mg + Tislelizumab 200 mg)
Number analyzed (Participants) | 24 | 28 | 44 | 26 | 17 | 18 | 0 | 39 | 54 | 22 | 19 | 22
percentage of participants
  ORR: TIGIT IC < 1%: number analyzed (Participants) | 0 | 0 | 0 | 12 | 0 | 0 | 0 | 0 | 0 | 9 | 12 | 9
  ORR: TIGIT IC < 1% |  |  |  | 58.3 [27.7 to 84.8] |  |  |  |  |  | 22.2 [2.8 to 60.0] | 16.7 [2.1 to 48.4] | 22.2 [2.8 to 60.0]
  ORR: TIGIT IC >= 1%: number analyzed (Participants) | 0 | 0 | 0 | 14 | 0 | 0 | 0 | 0 | 0 | 13 | 7 | 13
  ORR: TIGIT IC >= 1% |  |  |  | 57.1 [28.9 to 82.3] |  |  |  |  |  | 38.5 [13.9 to 68.4] | 42.9 [9.9 to 81.6] | 38.5 [13.9 to 68.4]
  ORR: TIGIT IC < 5%: number analyzed (Participants) | 11 | 15 | 17 | 0 | 9 | 8 | 0 | 11 | 25 | 0 | 0 | 0
  ORR: TIGIT IC < 5% | 54.5 [23.4 to 83.3] | 66.7 [38.4 to 88.2] | 17.6 [3.8 to 43.4] |  | 0.0 [0.0 to 33.6] | 62.5 [24.5 to 91.5] |  | 36.4 [10.9 to 69.2] | 56.0 [34.9 to 75.6] |  |  |
  ORR: TIGIT IC >= 5%: number analyzed (Participants) | 13 | 13 | 27 | 0 | 8 | 10 | 0 | 28 | 29 | 0 | 0 | 0
  ORR: TIGIT IC >= 5% | 61.5 [31.6 to 86.1] | 38.5 [13.9 to 68.4] | 55.6 [35.3 to 74.5] |  | 12.5 [0.3 to 52.7] | 70.0 [34.8 to 93.3] |  | 32.1 [15.9 to 52.4] | 44.8 [26.4 to 64.3] |  |  |

24. Secondary Outcome: Phase 1b (Cohort 1-10): Percentage of Participants With ORR: PD-L1 Biomarkers Expression
Description: Archival or fresh tumor samples were collected for analysis of biomarkers for T cell immunoglobulin and immunoreceptor tyrosine-based inhibitory motif (ITIM) domain (TIGIT) and PD-L1 expression.
  The PD-L1 expression scoring algorithm and the classification thresholds were also different for various cohorts as follows:
  For Cohort 1 and Cohort 2, PD-L1 TC <1% or >= 1%; for Cohorts 3, 5, and 10, PD-L1 TC < 50% or >=50%; for Cohort 4, PD-L1 tumor area positivity (TAP) <1% or >=1%; for Cohort 9, PD-L1 TAP < 5% or >= 5%; for Cohort 6 and 8, PD-L1 TAP <10% or >=10%. ORR is reported for each PD-L1 subgroup as relevant in each cohort. Biomarker data were not analyzed and reported for participants in Cohort 7.
Time Frame: Maximum time duration on study: up to 41.6 months (Cohorts 1 to 9) and up to 21.4 months (Cohort 10)
Population: Analysis was performed on efficacy evaluable analysis set for participants with available PD-L1 expression levels. Here, "Overall number of participants analyzed" = participants with available data for this outcome measure and "number analyzed" signifies participants with available data for each specified category at respective visit and "0" in the number analyzed defines no participant were available for analysis at specified time-points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1b: Dose Expansion: Cohort 1 | Phase 1b: Dose Expansion: Cohort 2 | Phase 1b: Dose Expansion: Cohort 3 | Phase 1b: Dose Expansion: Cohort 4 | Phase 1b: Dose Expansion: Cohort 5 | Phase 1b: Dose Expansion: Cohort 6 | Phase 1b: Dose Expansion: Cohort 7 | Phase 1b: Dose Expansion: Cohort 8 | Phase 1b: Dose Expansion: Cohort 9 | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 450 mg + Tislelizumab 200 mg) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 900 mg + Tislelizumab 200 mg) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 1800 mg + Tislelizumab 200 mg)
Number analyzed (Participants) | 25 | 29 | 45 | 24 | 17 | 17 | 0 | 37 | 55 | 23 | 19 | 23
percentage of participants
  ORR: PD-L1 TC < 1%: number analyzed (Participants) | 9 | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ORR: PD-L1 TC < 1% | 66.7 [29.9 to 92.5] | 60.0 [32.3 to 83.7] |  |  |  |  |  |  |  |  |  |
  ORR: PD-L1 TC >= 1%: number analyzed (Participants) | 16 | 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ORR: PD-L1 TC >= 1% | 56.3 [29.9 to 80.2] | 42.9 [17.7 to 71.1] |  |  |  |  |  |  |  |  |  |
  ORR: PD-L1 TC < 50%: number analyzed (Participants) | 0 | 0 | 26 | 0 | 12 | 0 | 0 | 0 | 0 | 15 | 11 | 15
  ORR: PD-L1 TC < 50% |  |  | 30.8 [14.3 to 51.8] |  | 0.0 [0.0 to 26.5] |  |  |  |  | 46.7 [21.3 to 73.4] | 18.2 [2.3 to 51.87] | 26.7 [7.8 to 55.1]
  ORR: PD-L1 TC >= 50%: number analyzed (Participants) | 0 | 0 | 19 | 0 | 5 | 0 | 0 | 0 | 0 | 8 | 8 | 8
  ORR: PD-L1 TC >= 50% |  |  | 52.6 [28.9 to 75.6] |  | 20.0 [0.5 to 71.6] |  |  |  |  | 12.5 [0.3 to 52.7] | 37.5 [8.5 to 75.5] | 50.0 [15.7 to 84.3]
  ORR: PD-L1 TAP < 1%: number analyzed (Participants) | 0 | 0 | 0 | 16 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ORR: PD-L1 TAP < 1% |  |  |  | 56.3 [29.9 to 80.2] |  |  |  |  |  |  |  |
  ORR: PD-L1 TAP >= 1%: number analyzed (Participants) | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ORR: PD-L1 TAP >= 1% |  |  |  | 50.0 [15.7 to 84.3] |  |  |  |  |  |  |  |
  ORR: PD-L1 TAP < 5%: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 28 | 0 | 0 | 0
  ORR: PD-L1 TAP < 5% |  |  |  |  |  |  |  |  | 50.0 [30.6 to 69.4] |  |  |
  ORR: PD-L1 TAP >= 5%: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 27 | 0 | 0 | 0
  ORR: PD-L1 TAP >= 5% |  |  |  |  |  |  |  |  | 55.6 [35.3 to 74.5] |  |  |
  ORR: PD-L1 TAP < 10%: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 13 | 0 | 16 | 0 | 0 | 0 | 0
  ORR: PD-L1 TAP < 10% |  |  |  |  |  | 61.5 [31.6 to 86.1] |  | 31.3 [11.0 to 58.7] |  |  |  |
  ORR: PD-L1 TAP >= 10%: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 21 | 0 | 0 | 0 | 0
  ORR: PD-L1 TAP >= 10% |  |  |  |  |  | 100.0 [39.8 to 100.0] |  | 38.1 [18.1 to 61.6] |  |  |  |

25. Secondary Outcome: Phase 1b (Cohort 1-10): PFS in TIGIT Biomarkers Expression
Description: Archival or fresh tumor samples were collected for analysis of biomarkers for T cell immunoglobulin and immunoreceptor tyrosine-based inhibitory motif (ITIM) domain (TIGIT) and PD-L1 expression.
  The TIGIT expression on immune cells and the classification thresholds were different for various cohorts. For Cohort 4, TIGIT IC was categorized as <1% or >=1%; for Cohorts 1, 2, 3, 5, 6, 8, 9 and 10, TIGIT IC was categorized as <5% or >=5%. Median PFS (mPFS) is reported for each TIGIT subgroup as relevant in each cohort. Biomarker data were not analyzed and reported for participants in Cohort 7.
Time Frame: Maximum time duration on study: up to 41.6 months (Cohorts 1 to 9) and up to 21.4 months (Cohort 10)
Population: Analysis was performed on efficacy evaluable analysis set. Here, "Overall number of participants analyzed" = participants with available data for this outcome measure and "number analyzed" signifies participants with available data for each specified category at respective visit and "0" in the number analyzed defines no participant were available for analysis at specified time-points.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b: Dose Expansion: Cohort 1 | Phase 1b: Dose Expansion: Cohort 2 | Phase 1b: Dose Expansion: Cohort 3 | Phase 1b: Dose Expansion: Cohort 4 | Phase 1b: Dose Expansion: Cohort 5 | Phase 1b: Dose Expansion: Cohort 6 | Phase 1b: Dose Expansion: Cohort 7 | Phase 1b: Dose Expansion: Cohort 8 | Phase 1b: Dose Expansion: Cohort 9 | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 450 mg + Tislelizumab 200 mg) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 900 mg + Tislelizumab 200 mg) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 1800 mg + Tislelizumab 200 mg)
Number analyzed (Participants) | 25 | 29 | 44 | 27 | 17 | 19 | 0 | 41 | 55 | 23 | 21 | 22
months
  mPFS: TIGIT IC < 1%: number analyzed (Participants) | 0 | 0 | 0 | 13 | 0 | 0 | 0 | 0 | 0 | 9 | 13 | 9
  mPFS: TIGIT IC < 1% |  |  |  | 5.1 [1.2 to 5.6] |  |  |  |  |  | 2.7 [1.2 to 6.9] | 1.6 [1.2 to 6.9] | 5.5 [1.4 to 9.5]
  mPFS: TIGIT IC >= 1%: number analyzed (Participants) | 0 | 0 | 0 | 14 | 0 | 0 | 0 | 0 | 0 | 14 | 8 | 13
  mPFS: TIGIT IC >= 1% |  |  |  | 4.9 [4.1 to 7.4] |  |  |  |  |  | 2.8 [1.3 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 9.0 [0.6 to 12.3] | 8.5 [5.7 to 11.6]
  mPFS: TIGIT IC < 5%: number analyzed (Participants) | 12 | 15 | 17 | 0 | 9 | 9 | 0 | 12 | 25 | 0 | 0 | 0
  mPFS: TIGIT IC < 5% | 7.0 [3.4 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 10.9 [5.3 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 5.4 [2.6 to 15.0] |  | 3.8 [1.2 to 5.3] | 8.1 [0.4 to 12.3] |  | 6.1 [4.0 to 12.5] | 6.9 [4.1 to 11.1] |  |  |
  mPFS: TIGIT IC >= 5%: number analyzed (Participants) | 13 | 14 | 27 | 0 | 8 | 10 | 0 | 29 | 30 | 0 | 0 | 0
  mPFS: TIGIT IC >= 5% | 6.9 [3.9 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 12.6 [5.4 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 5.5 [4.2 to 11.0] |  | 5.2 [1.0 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 7.9 [3.0 to 12.2] |  | 4.1 [1.4 to 8.3] | 8.2 [2.8 to 11.2] |  |  |

26. Secondary Outcome: Phase 1b (Cohort 1-10): PFS in PD-L1 Biomarkers Expression
Description: Archival or fresh tumor samples were collected for analysis of biomarkers for T cell immunoglobulin and immunoreceptor tyrosine-based inhibitory motif (ITIM) domain (TIGIT) and PD-L1 expression. The PD-L1 expression scoring algorithm and the classification thresholds were also different for various cohorts as follows:
  For Cohort 1 and Cohort 2, PD-L1 TC <1% or >= 1%; for Cohorts 3, 5, and 10, PD-L1 TC < 50% or >=50%; for Cohort 4, PD-L1 tumor area positivity (TAP) <1% or >=1%; for Cohort 9, PD-L1 TAP < 5% or >= 5%; for Cohort 6 and 8, PD-L1 TAP <10% or >=10%. mPFS is reported for each PD-L1 subgroup as relevant in each cohort. Biomarker data were not analyzed and reported for participants in Cohort 7.
Time Frame: Maximum time duration on study: up to 41.6 months (Cohorts 1 to 9) and up to 21.4 months (Cohort 10)
Population: as for outcome 25
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b: Dose Expansion: Cohort 1 | Phase 1b: Dose Expansion: Cohort 2 | Phase 1b: Dose Expansion: Cohort 3 | Phase 1b: Dose Expansion: Cohort 4 | Phase 1b: Dose Expansion: Cohort 5 | Phase 1b: Dose Expansion: Cohort 6 | Phase 1b: Dose Expansion: Cohort 7 | Phase 1b: Dose Expansion: Cohort 8 | Phase 1b: Dose Expansion: Cohort 9 | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 450 mg + Tislelizumab 200 mg) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 900 mg + Tislelizumab 200 mg) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 1800 mg + Tislelizumab 200 mg)
Number analyzed (Participants) | 26 | 30 | 45 | 25 | 17 | 18 | 0 | 39 | 56 | 24 | 21 | 23
months
  mPFS: PD-L1 TC < 1%: number analyzed (Participants) | 9 | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  mPFS: PD-L1 TC < 1% | 7.0 [0.3 to NA] — Upper limit of 95% CI could not be calculated due to an insufficient number of participants with events. | 23.6 [5.4 to NA] — Upper limit of 95% CI could not be calculated due to an insufficient number of participants with events. |  |  |  |  |  |  |  |  |  |
  mPFS: PD-L1 TC >= 1%: number analyzed (Participants) | 17 | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  mPFS: PD-L1 TC >= 1% | 6.9 [5.4 to NA] — Upper limit of 95% CI could not be calculated due to an insufficient number of participants with events. | 8.0 [6.3 to 16.5] |  |  |  |  |  |  |  |  |  |
  mPFS: PD-L1 TC < 50%: number analyzed (Participants) | 0 | 0 | 26 | 0 | 12 | 0 | 0 | 0 | 0 | 16 | 13 | 15
  mPFS: PD-L1 TC < 50% |  |  | 5.2 [3.0 to 5.5] |  | 1.6 [1.2 to 5.0] |  |  |  |  | 6.4 [1.2 to NA] — Upper limit of 95% CI could not be calculated due to an insufficient number of participants with events. | 1.4 [1.1 to 6.9] | 8.5 [4.2 to 11.6]
  mPFS: PD-L1 TC >= 50%: number analyzed (Participants) | 0 | 0 | 19 | 0 | 5 | 0 | 0 | 0 | 0 | 8 | 8 | 8
  mPFS: PD-L1 TC >= 50% |  |  | 8.2 [4.2 to 23.9] |  | 20.6 [1.4 to NA] — Upper limit of 95% CI could not be calculated due to an insufficient number of participants with events. |  |  |  |  | 2.6 [1.3 to 5.5] | 9.0 [0.6 to 12.3] | 6.8 [1.4 to NA] — Upper limit of 95% CI could not be calculated due to an insufficient number of participants with events.
  mPFS: PD-L1 TAP < 1%: number analyzed (Participants) | 0 | 0 | 0 | 17 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  mPFS: PD-L1 TAP < 1% |  |  |  | 5.1 [4.1 to 5.6] |  |  |  |  |  |  |  |
  mPFS: PD-L1 TAP >= 1%: number analyzed (Participants) | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  mPFS: PD-L1 TAP >= 1% |  |  |  | 5.4 [0.7 to 7.4] |  |  |  |  |  |  |  |
  mPFS: PD-L1 TAP < 5%: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 28 | 0 | 0 | 0
  mPFS: PD-L1 TAP < 5% |  |  |  |  |  |  |  |  | 6.7 [2.8 to 9.1] |  |  |
  mPFS: PD-L1 TAP >= 5%: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 28 | 0 | 0 | 0
  mPFS: PD-L1 TAP >= 5% |  |  |  |  |  |  |  |  | 8.2 [3.9 to 11.1] |  |  |
  mPFS: PD-L1 TAP < 10%: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 13 | 0 | 18 | 0 | 0 | 0 | 0
  mPFS: PD-L1 TAP < 10% |  |  |  |  |  | 7.6 [3.7 to 10.7] |  | 4.0 [1.2 to 12.4] |  |  |  |
  mPFS: PD-L1 TAP >= 10%: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 21 | 0 | 0 | 0 | 0
  mPFS: PD-L1 TAP >= 10% |  |  |  |  |  | 10.3 [2.7 to NA] — Upper limit of 95% CI could not be calculated due to an insufficient number of participants with events. |  | 7.1 [3.0 to 9.7] |  |  |  |

ADVERSE EVENTS:
Time Frame: All cause-mortality data was collected from randomization through end of study (up to 5 years). SAEs & non-serious AEs data: up to 30 days after last dose of study drugs (Maximum time duration on study: up to 35.7 months (escalation cohort); up to 13.3 months (verification cohort); up to 41.6 months [Cohorts 1 to 9] & up to 21.4 months [Cohort 10])
Description: Analysis was performed on safety set.
Groups:
- Phase 1: Dose Escalation: Ociperlimab 50 mg + Tislelizumab 200 mg: Participants received ociperlimab 50 mg IV infusion on Day 1 of each cycle (cycle 1= 28 days) and tislelizumab 200 mg IV infusion on Day 8 of Cycle 1. If tolerated, participants received ociperlimab and tislelizumab IV on Cycle 2 Day 1 (cycle 2 onwards = 21 days) and thereafter every 21 days (i.e., Q3W) until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
- Phase 1: Dose Escalation: Ociperlimab 150 mg + Tislelizumab 200 mg: Participants received ociperlimab 150 mg IV infusion on Day 1 of each cycle (cycle 1= 28 days) and tislelizumab 200 mg IV infusion on Day 8 of Cycle 1. If tolerated, participants received ociperlimab and tislelizumab IV on Cycle 2 Day 1 (cycle 2 onwards = 21 days) and thereafter every 21 days (i.e. Q3W) until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
- Phase 1: Dose Escalation: Ociperlimab 450 mg + Tislelizumab 200 mg: Participants received ociperlimab 450 mg IV infusion on Day 1 of each cycle (cycle 1= 28 days) and tislelizumab 200 mg IV infusion on Day 8 of Cycle 1. If tolerated, participants received ociperlimab and tislelizumab IV on Cycle 2 Day 1 (cycle 2 onwards = 21 days) and thereafter every 21 days (i.e. Q3W) until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
- Phase 1: Dose Escalation: Ociperlimab 900 mg + Tislelizumab 200 mg: Participants received ociperlimab 900 mg IV infusion on Day 1 of each cycle (cycle 1= 28 days) and tislelizumab 200 mg IV infusion on Day 8 of Cycle 1. If tolerated, participants received ociperlimab and tislelizumab IV on Cycle 2 Day 1 (cycle 2 onwards = 21 days) and thereafter every 21 days (i.e. Q3W) until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
- Phase 1: Dose Escalation: Ociperlimab 1800 mg + Tislelizumab 200 mg: Participants received ociperlimab 1800 mg IV infusion on Day 1 of each cycle (cycle 1= 28 days) and tislelizumab 200 mg IV infusion on Day 8 of Cycle 1. If tolerated, participants received ociperlimab and tislelizumab IV on Cycle 2 Day 1 (cycle 2 onwards = 21 days) and thereafter every 21 days (i.e. Q3W) until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
- Phase 1: Dose Verification: Cohort 1A (Ociperlimab 900 mg): Participants received ociperlimab 900 mg as monotherapy as IV infusion on Day 1 of each 21-day treatment cycle and will be followed up until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
- Phase 1: Dose Verification: Cohort 1B (Ociperlimab 900 mg + Tislelizumab 200 mg): Participants received ociperlimab 900 mg as IV infusion on Day 1 of each 21-day treatment cycle and tislelizumab 200 mg IV infusion once every 21 days (i.e. Q3W) until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
- Phase 1b: Dose Expansion: Cohort 1: Participants with metastatic squamous NSCLC received treatment with ociperlimab 900 mg IV infusion along with tislelizumab 200 mg IV infusion on Day 1 of each 21-day cycle. Participants also received 4 to 6 cycles of chemo with carboplatin AUC 5 or 6 (Day 1) + paclitaxel 200 or 175 mg/m^2 (Day 1) or nab paclitaxel 100 mg/m^2 (Days 1, 8 and 15) Q3W and were followed up until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
- Phase 1b: Dose Expansion: Cohort 2: Participants with metastatic NSCLC (PD-L1 positive, TC>= 1%) received treatment with ociperlimab 900 mg IV infusion and tislelizumab 200 mg IV infusion on Day 1 of each 21-day cycle. Participants also received cisplatin 75 mg/m^2 or carboplatin (AUC 5) and pemetrexed 500 mg/m^2 (on Day 1) Q3W for 4-6 cycles followed by ociperlimab 900 mg + tislelizumab 200 mg + pemetrexed 500 mg/m^2 on Day 1 Q3W and were followed up until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
- Phase 1b: Dose Expansion: Cohort 3: Participants with metastatic NSCLC (PD-L1 positive, TC >=1%) were treated with ociperlimab 900 mg IV infusion and tislelizumab 200 mg IV infusion on Day 1 of each 21-day cycle and were followed up until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
- Phase 1b: Dose Expansion: Cohort 4: Participants with extensive-stage SCLC received treatment with ociperlimab 900 mg IV infusion, tislelizumab 200 mg IV infusion. Participants also received 4 cycles of etoposide 100 mg/m^2 (on Days 1, 2, 3), and cisplatin 75 mg/m^2 /carboplatin AUC 5 (Day 1) Q3W, followed by ociperlimab 900 mg (Day 1) + tislelizumab 200 mg (Day 1) Q3W and were followed up until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
- Phase 1b: Dose Expansion: Cohort 5: Checkpoint inhibitor (CPI)-experienced NSCLC participants received treatment with ociperlimab 900 mg IV infusion and tislelizumab 200 mg IV infusions on Day 1 of each 21-day cycle and were followed up until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
- Phase 1b: Dose Expansion: Cohort 7: Participants with metastatic EAC received treatment with 6 cycles of ociperlimab 900 mg (Day 1) IV infusion, tislelizumab 200 mg (Day 1) IV infusion, cisplatin 75 mg/m^2 (Day 1), and Fluorouracil 750-800 mg/m^2 (5-FU; Day 1 to Day 5) or paclitaxel 200 or 175 mg/m^2 (Day 1) Q3W followed by ociperlimab 900 mg and tislelizumab 200 mg on Day 1 of every 21-day cycle and were followed up until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
- Phase 1b: Dose Expansion: Cohort 8: Participants with recurrent or metastatic head and neck squamous cell carcinoma (HNSCC; PD-L1 positive, vCPS >= 1%) received treatment with ociperlimab 900 mg IV infusion and tislelizumab 200 mg IV infusions on Day 1 of every 21-day cycle and were followed up until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
- Phase 1b: Dose Expansion: Cohort 9: Participants with unresectable, locally advanced, recurrent, or metastatic G/GEJ adenocarcinoma received treatment with 6 cycles of ociperlimab 900 mg (Day 1) IV infusion, tislelizumab 200 mg (Day 1) IV infusion, (oxaliplatin 1300 mg/m^2 [Day 1] and capecitabine 1000 mg/m^2 [Day 1-14 twice daily], or cisplatin 75 mg/m^2 [Day], and 5-FU 750-800 mg/m^2 [Day 1-5]) Q3W followed by ociperlimab 900 mg (Day 1), tislelizumab 200 mg (Day 1) + capecitabine 1000 mg/m^2 twice daily (Day 1-14) Q3W and were followed up until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
- Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 1800 mg + Tislelizumab 200 mg): Participants with metastatic NSCLC (PD-L1 positive, TC >= 1%) received treatment with ociperlimab 1800 mg IV infusion and tislelizumab 200 mg IV infusion on Day 1 of every 21-day cycle and were followed up until disease progression, AEs, participant withdrew consent, lost to follow-up or death, whichever came first.
Arm/Group | Phase 1: Dose Escalation: Ociperlimab 50 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 150 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 450 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 900 mg + Tislelizumab 200 mg | Phase 1: Dose Escalation: Ociperlimab 1800 mg + Tislelizumab 200 mg | Phase 1: Dose Verification: Cohort 1A (Ociperlimab 900 mg) | Phase 1: Dose Verification: Cohort 1B (Ociperlimab 900 mg + Tislelizumab 200 mg) | Phase 1b: Dose Expansion: Cohort 1 | Phase 1b: Dose Expansion: Cohort 2 | Phase 1b: Dose Expansion: Cohort 3 | Phase 1b: Dose Expansion: Cohort 4 | Phase 1b: Dose Expansion: Cohort 5 | Phase 1b: Dose Expansion: Cohort 6 | Phase 1b: Dose Expansion: Cohort 7 | Phase 1b: Dose Expansion: Cohort 8 | Phase 1b: Dose Expansion: Cohort 9 | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 900 mg + Tislelizumab 200 mg) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 450 mg + Tislelizumab 200 mg) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 1800 mg + Tislelizumab 200 mg)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/3 | 4/6 | 7/16 | 2/6 | 4/9 | 3/11 | 24/41 | 24/43 | 22/45 | 35/43 | 18/26 | 14/21 | 6/6 | 19/41 | 42/60 | 8/21 | 9/24 | 10/23
Serious Adverse Events (participants affected / at risk) | 1/1 | 2/3 | 3/6 | 9/16 | 1/6 | 3/9 | 5/11 | 21/41 | 28/43 | 15/45 | 23/43 | 9/26 | 11/21 | 4/6 | 22/41 | 32/60 | 8/21 | 10/24 | 13/23
Other Adverse Events (participants affected / at risk) | 1/1 | 3/3 | 6/6 | 13/16 | 6/6 | 8/9 | 11/11 | 40/41 | 42/43 | 44/45 | 41/43 | 24/26 | 21/21 | 6/6 | 39/41 | 59/60 | 17/21 | 22/24 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Dose Escalation: Ociperlimab 50 mg + Tislelizumab 200 mg (N=1) | Phase 1: Dose Escalation: Ociperlimab 150 mg + Tislelizumab 200 mg (N=3) | Phase 1: Dose Escalation: Ociperlimab 450 mg + Tislelizumab 200 mg (N=6) | Phase 1: Dose Escalation: Ociperlimab 900 mg + Tislelizumab 200 mg (N=16) | Phase 1: Dose Escalation: Ociperlimab 1800 mg + Tislelizumab 200 mg (N=6) | Phase 1: Dose Verification: Cohort 1A (Ociperlimab 900 mg) (N=9) | Phase 1: Dose Verification: Cohort 1B (Ociperlimab 900 mg + Tislelizumab 200 mg) (N=11) | Phase 1b: Dose Expansion: Cohort 1 (N=41) | Phase 1b: Dose Expansion: Cohort 2 (N=43) | Phase 1b: Dose Expansion: Cohort 3 (N=45) | Phase 1b: Dose Expansion: Cohort 4 (N=43) | Phase 1b: Dose Expansion: Cohort 5 (N=26) | Phase 1b: Dose Expansion: Cohort 6 (N=21) | Phase 1b: Dose Expansion: Cohort 7 (N=6) | Phase 1b: Dose Expansion: Cohort 8 (N=41) | Phase 1b: Dose Expansion: Cohort 9 (N=60) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 900 mg + Tislelizumab 200 mg) (N=21) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 450 mg + Tislelizumab 200 mg) (N=24) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 1800 mg + Tislelizumab 200 mg) (N=23)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nodal rhythm (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Primary adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 6 (6) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 8 (10) | 1 (1) | 0 (0) | 1 (1) | 3 (4)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shoulder fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Human rhinovirus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somatic dysfunction (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid sinus syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalitis autoimmune (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bipolar I disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Embolism venous (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Dose Escalation: Ociperlimab 50 mg + Tislelizumab 200 mg (N=1) | Phase 1: Dose Escalation: Ociperlimab 150 mg + Tislelizumab 200 mg (N=3) | Phase 1: Dose Escalation: Ociperlimab 450 mg + Tislelizumab 200 mg (N=6) | Phase 1: Dose Escalation: Ociperlimab 900 mg + Tislelizumab 200 mg (N=16) | Phase 1: Dose Escalation: Ociperlimab 1800 mg + Tislelizumab 200 mg (N=6) | Phase 1: Dose Verification: Cohort 1A (Ociperlimab 900 mg) (N=9) | Phase 1: Dose Verification: Cohort 1B (Ociperlimab 900 mg + Tislelizumab 200 mg) (N=11) | Phase 1b: Dose Expansion: Cohort 1 (N=41) | Phase 1b: Dose Expansion: Cohort 2 (N=43) | Phase 1b: Dose Expansion: Cohort 3 (N=45) | Phase 1b: Dose Expansion: Cohort 4 (N=43) | Phase 1b: Dose Expansion: Cohort 5 (N=26) | Phase 1b: Dose Expansion: Cohort 6 (N=21) | Phase 1b: Dose Expansion: Cohort 7 (N=6) | Phase 1b: Dose Expansion: Cohort 8 (N=41) | Phase 1b: Dose Expansion: Cohort 9 (N=60) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 900 mg + Tislelizumab 200 mg) (N=21) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 450 mg + Tislelizumab 200 mg) (N=24) | Phase 1b: Dose Optimization: Cohort 10: (Ociperlimab 1800 mg + Tislelizumab 200 mg) (N=23)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 2 (3) | 15 (38) | 30 (95) | 8 (9) | 24 (42) | 3 (3) | 14 (27) | 1 (1) | 5 (7) | 30 (45) | 5 (6) | 4 (5) | 7 (12)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (8) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 1 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 0 (0) | 0 (0) | 0 (0)
Atrial escape rhythm (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 1 (1) | 2 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Hypopituitarism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 5 (5) | 4 (4) | 7 (8) | 0 (0) | 4 (6) | 1 (1) | 9 (10) | 13 (18) | 0 (0) | 1 (1) | 3 (5)
Thyroid disorder (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Night blindness (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papilloedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal drusen (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulcerative keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 3 (5) | 2 (2) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (2)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal pruritus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 11 (12) | 10 (16) | 3 (3) | 12 (17) | 2 (2) | 7 (9) | 3 (3) | 9 (9) | 9 (16) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 3 (4) | 7 (10) | 5 (12) | 7 (10) | 3 (4) | 5 (8) | 1 (1) | 4 (5) | 13 (18) | 1 (1) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (6) | 0 (0) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eosinophilic oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal mucosal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip blister (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 9 (12) | 12 (40) | 11 (14) | 8 (13) | 2 (2) | 8 (13) | 2 (2) | 3 (3) | 24 (47) | 3 (3) | 1 (1) | 3 (3)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Parotid gland enlargement (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Poor dental condition (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary gland pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 3 (4) | 1 (3) | 3 (4) | 2 (2) | 2 (2) | 10 (17) | 1 (1) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 6 (8) | 4 (4) | 6 (8) | 2 (2) | 3 (5) | 2 (3) | 3 (3) | 15 (28) | 2 (2) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 7 (17) | 6 (6) | 2 (2) | 6 (9) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 7 (7) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 8 (11) | 2 (2) | 3 (3) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 4 (5) | 3 (4) | 2 (2) | 0 (0) | 2 (2) | 4 (4) | 8 (9) | 6 (10) | 4 (4) | 8 (9) | 3 (5) | 4 (6) | 5 (6) | 17 (26) | 1 (2) | 0 (0) | 3 (3)
Feeling of body temperature change (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 7 (9) | 4 (6) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 9 (14) | 3 (3) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 6 (8) | 4 (5) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 3 (3) | 9 (13) | 4 (5) | 13 (14) | 4 (5) | 0 (0) | 4 (4) | 1 (1) | 3 (3) | 12 (17) | 3 (3) | 5 (7) | 3 (6)
Temperature intolerance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 2 (2) | 2 (2) | 1 (2) | 6 (9) | 0 (0) | 1 (1) | 8 (9) | 0 (0) | 1 (1) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatophytosis of nail (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mediastinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 5 (5) | 4 (4) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 4 (4) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (3) | 7 (8) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (3) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stoma site discharge (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 10 (14) | 15 (37) | 8 (10) | 5 (7) | 0 (0) | 6 (7) | 0 (0) | 4 (6) | 8 (16) | 0 (0) | 4 (4) | 3 (3)
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 3 (7) | 5 (7) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 5 (9) | 0 (0) | 0 (0) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (5) | 10 (13) | 15 (35) | 8 (11) | 6 (6) | 0 (0) | 5 (5) | 0 (0) | 4 (5) | 12 (21) | 0 (0) | 2 (2) | 4 (4)
Beta 2 microglobulin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bile acids increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bilirubin conjugated increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 5 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (2) | 0 (0) | 1 (1)
Bilirubin urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (4) | 3 (4) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 3 (4) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 3 (4) | 3 (7) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 3 (3) | 5 (9) | 2 (2) | 0 (0) | 1 (1)
Blood bilirubin unconjugated increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood chloride decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Blood cholinesterase decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase MB increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 2 (5) | 2 (2) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 2 (5) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 2 (3) | 3 (5) | 1 (2) | 2 (2) | 7 (16) | 2 (3) | 3 (3) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (2) | 7 (19) | 2 (2) | 3 (6) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 6 (13) | 2 (3) | 1 (1) | 2 (5)
Blood phosphorus increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood testosterone decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (8) | 1 (1) | 1 (1) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain natriuretic peptide increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 5 (14) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (5) | 0 (0) | 1 (2)
Electrocardiogram T wave abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibrin D dimer increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Fibrinogen degradation products increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 5 (10) | 1 (1) | 5 (7) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Glucose urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glutathione reductase activity increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glycocholic acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 4 (5) | 5 (6) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 6 (8) | 2 (2) | 1 (1) | 6 (9)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (6) | 3 (14) | 0 (0) | 4 (12) | 0 (0) | 2 (4) | 1 (1) | 2 (2) | 5 (6) | 0 (0) | 1 (1) | 1 (2)
Myoglobin blood increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 18 (59) | 19 (89) | 1 (1) | 23 (51) | 1 (1) | 11 (28) | 1 (1) | 1 (1) | 20 (94) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Occult blood positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 12 (33) | 14 (26) | 1 (2) | 12 (21) | 0 (0) | 7 (11) | 0 (0) | 1 (1) | 24 (68) | 1 (1) | 0 (0) | 1 (1)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Protein total decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (3) | 0 (0)
Protein urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Red blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Red blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Thyroxine decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroxine free decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroxine free increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tri-iodothyronine decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tri-iodothyronine free increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Urobilinogen urine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin D decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (4) | 2 (2) | 5 (6) | 3 (3) | 2 (2) | 4 (4) | 5 (5) | 3 (4) | 1 (2) | 4 (4) | 13 (13) | 2 (2) | 1 (1) | 5 (5)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 6 (7) | 3 (3) | 0 (0) | 3 (4) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 15 (66) | 18 (98) | 0 (0) | 16 (36) | 0 (0) | 14 (41) | 0 (0) | 0 (0) | 19 (101) | 0 (0) | 1 (2) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 3 (4) | 15 (35) | 14 (19) | 9 (10) | 2 (2) | 5 (6) | 5 (8) | 0 (0) | 2 (2) | 17 (33) | 4 (6) | 2 (2) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 2 (3) | 2 (3) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 5 (9) | 0 (0) | 1 (1) | 0 (0)
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 4 (6) | 5 (16) | 5 (18) | 3 (3) | 2 (5) | 0 (0) | 3 (5) | 0 (0) | 1 (1) | 3 (5) | 0 (0) | 2 (4) | 2 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 1 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (8) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (5) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 1 (2) | 5 (19) | 2 (2) | 2 (4) | 0 (0) | 4 (10) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 7 (13) | 6 (18) | 4 (6) | 4 (10) | 0 (0) | 6 (15) | 0 (0) | 10 (11) | 14 (32) | 2 (3) | 5 (5) | 9 (12)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 10 (18) | 0 (0) | 0 (0) | 3 (7)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (4) | 4 (6) | 3 (6) | 6 (6) | 1 (1) | 5 (6) | 1 (1) | 2 (3) | 8 (16) | 2 (2) | 3 (3) | 1 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 7 (10) | 0 (0) | 0 (0) | 4 (8) | 0 (0) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 5 (6) | 8 (20) | 2 (2) | 6 (10) | 1 (2) | 6 (10) | 0 (0) | 8 (11) | 16 (26) | 3 (3) | 2 (3) | 3 (7)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 4 (6) | 1 (1) | 0 (0) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 3 (5) | 2 (2) | 0 (0) | 0 (0) | 7 (12) | 5 (14) | 4 (4) | 5 (5) | 3 (5) | 2 (3) | 0 (0) | 4 (4) | 2 (2) | 1 (1) | 3 (4) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 8 (8) | 8 (9) | 1 (1) | 3 (4) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (6) | 3 (3) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 5 (8) | 3 (3) | 4 (7) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemangioma of spleen (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Akathisia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain fog (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 3 (4) | 5 (5) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 3 (4) | 6 (12) | 2 (2) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 2 (2) | 3 (4) | 1 (1) | 1 (1) | 2 (2) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 7 (11) | 1 (4) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Paraparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 19 (31) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fear of falling (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Frigophobia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (7) | 1 (1) | 5 (5) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 5 (8) | 2 (2) | 1 (1) | 2 (2)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 1 (2)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Ureteric dilatation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 6 (6) | 5 (5) | 7 (7) | 5 (7) | 7 (7) | 2 (3) | 0 (0) | 2 (2) | 2 (6) | 0 (0) | 6 (6) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 7 (8) | 6 (8) | 5 (5) | 3 (4) | 2 (2) | 0 (0) | 1 (1) | 4 (5) | 3 (5) | 2 (2) | 4 (4) | 2 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 4 (4) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paranasal sinus inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 6 (7) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 5 (5)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 14 (14) | 2 (3) | 0 (0) | 5 (5) | 1 (1) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 1 (1) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 13 (20) | 0 (0) | 0 (0) | 0 (0)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 18 (24) | 10 (13) | 17 (29) | 9 (15) | 4 (6) | 5 (5) | 1 (1) | 11 (15) | 13 (19) | 2 (2) | 3 (4) | 7 (10)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 2 (2) | 2 (3) | 15 (36) | 18 (28) | 11 (19) | 8 (8) | 6 (6) | 7 (9) | 0 (0) | 9 (10) | 12 (15) | 2 (3) | 5 (5) | 5 (5)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 5 (6) | 2 (3) | 1 (2) | 0 (0) | 1 (1) | 2 (3) | 4 (9) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Superficial inflammatory dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Embolism venous (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (2) | 0 (0) | 1 (4) | 0 (0) | 2 (2) | 3 (5) | 1 (1) | 1 (1) | 5 (17) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Jugular vein embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Penetrating aortic ulcer (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scalp haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2023-11-10): https://cdn.clinicaltrials.gov/large-docs/62/NCT04047862/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-27): https://cdn.clinicaltrials.gov/large-docs/62/NCT04047862/SAP_001.pdf